Optimize PRO Study

NCT: 04091048

Study Protocol/Document Date: 20Sep2019

Version 4.0




| Medtronic Clinical Investigation Plan | |
|---|---|
| Study Product Name | Medtronic Evolut™ PRO System and Medtronic Evolut™ PRO+ System |
| Sponsor/Local Sponsor | Medtronic, Inc. Coronary and Structural Heart Clinical |
| | Medtronic of Canada Ltd. |
| Document Version | 4.0, 20 SEP 2019 |
| Co-Principal Investigators | Dr. Kendra Grubb<br>Emory University Hospital |
| | Dr. Steven Yakubov<br>Riverside Methodist Hospital / Ohio Health Research<br>Institute |
| Cor | nfidentiality Statement |
| he information contained in this docume | ent is confidential and the proprietary property of Medtron |

The information contained in this document is confidential and the proprietary property of Medtronic. Any distribution, copying, or disclosure without the prior written authorization of Medtronic is strictly prohibited. Persons to whom the information is disclosed must know that it is confidential and that it may not be further disclosed by them.




## 1. Investigator Statement

| Study product Name | Medtronic Evolut™ PRO and Medtronic Evolut™ PRO+ |
|---------------------|--------------------------------------------------|
| Sponsor | Medtronic Coronary and Structural Heart Clinical |
| Version Number/Date | 4.0, 20 September 2019 |

I have read the protocol, including all appendices, and I agree that it contains all necessary details for me and my staff to conduct this study as described. I will conduct this study as outlined herein and will make a reasonable effort to complete the study within the time designated.

I agree to comply with local and internal institutional requirements including the protocol, GCP, and ethical principles that have their origin in the Declaration of Helsinki.

I agree to ensure that the confidential information contained in this document will not be used for any purpose other than the evaluation and conduct of the clinical study without the prior written consent of Medtronic.

I will provide all study personnel under my supervision copies of the protocol and access to all information provided by Medtronic. I will discuss this material with them to ensure that they are fully informed about the products and the study.

| Investigator's Signature: |
|---------------------------|
| Investigator's Name: |
| Institution: |
| Date: |


## **Table of Contents**

| 1. | Investi | gator Statement | 2 |
|-----|-----------|-----------------------------------------------------|----|
| Tab | le of Co | ntents | 3 |
| 2. | Glossa | ry | 8 |
| 3. | Synops | sis | 10 |
| 4. | Introd | uction | 17 |
| 4 | .1. Back | ground and Rationale | 12 |
| 4 | .2. Purp | oose | 13 |
| 5. | Object | ives and Endpoints | 13 |
| 5 | .1. Obje | ectives | 13 |
| | 5.1.1. | Primary Objective | 13 |
| 5 | .2. Endp | ooints | 13 |
| | 5.2.1. | Primary Endpoint | 13 |
| | 5.2.2. | Secondary Endpoints | 13 |
| | 5.2.3. | Additional Exploratory Endpoints | 14 |
| | 5.2.4. | Rationale | 14 |
| 6. | Study I | Design | 14 |
| 6 | .1. Dura | ation | 14 |
| 6 | .2. Trial | Organization | 15 |
| | 6.2.1 | Participating Sites | 15 |
| | 6.2.2. | Site Principal Investigator | |
| | 6.2.2 | Heart Team | 15 |
| | 6.2.3 | Publication Committee | 15 |
| | 6.2.4 | Trial Training | 16 |
| 7. | Produc | t Description | 16 |
| 7 | | cription of Devices | |
| | | '<br>∕ledtronic Evolut PRO and Evolut™ PRO+ Systems | |
| 7 | | rufacturer | |
| 7 | .3. Intei | nded Population | 24 |

| 1/0 | rcian | |
|-----|-------|-----|
| ve | rsion | 4.0 |

#### 

| | 7.4. Prod | duct Training Requirements | 24 |
|---|---|---|---|
| | 7.5. Prod | duct Labeling, Tracking, and Accountability | 24 |
| | 7.6. Prod | duct Storage | 25 |
| 8. | Selecti | on of Subjects | 25 |
| | 8.1 Stud | ly Population | 25 |
| | 8.2. Subj | ect Enrollment | 25 |
| | 8.2.2. | Roll-In Subjects | 25 |
| | 8.3. Inclu | usion Criteria | 25 |
| | 8.4. Excl | usion Criteria | 26 |
| 9. | Study | Procedures | 27 |
| | 9.1 Sche | edule of Events | 27 |
| | 9.1.1 | Screening Procedures | 27 |
| | 9.1.2 | Enrollment | 28 |
| | 9.1.3 | Implant Procedure (TAVR) | 28 |
| | 9.1.3.1 | Procedural Angiogram | 29 |
| | 9.1.4 | Prior to Discharge | 30 |
| | 9.1.5 | Follow-Up Evaluations | 30 |
| | 9.1.6 | Additional Evaluations for Pacemaker Implants | 32 |
| | 9.1.7 | Missed Follow-Up Visits | 32 |
| | 9.1.8 | Core Labs | 32 |
| | 9.1.9 | Informed Consent | 32 |
| | 9.2 Revi | sions in Patient Information and Informed Consent Form | 33 |
| | 9.3 Asse | essment of Efficacy | 33 |
| | 9.4 Asse | essment of Safety | 33 |
| | 9.4.1 | Adverse Events and Device Deficiencies | 3 |
| | 9.5 Devi | ce Malfunction or Explant | 34 |
| | 9.6 Reco | ording Data | 34 |
| | 9.6.1 | Source Documents | 3 |
| | 9.7 Devi | ation Handling | 36 |


| | 9.8 Subj | ject Withdrawal or Discontinuation | 36 |
|---|---|---|---|
| 10 | Risks a | and Benefits | 37 |
| | 10.1 Pote | ential Risks | 37 |
| | 10.2 Pote | ential Benefits | 37 |
| | 10.3 Risk | -Benefit Rationale | 37 |
| | 10.3.1 | Measures to Mitigate Risks in the Trial Subjects | 37 |
| | 10.3.2 | Alternatives | 37 |
| | 10.3.3 | Results from the Risk Analysis and Justification for the Study | 38 |
| 11 | . Advers | se Events and Device Deficiencies | 38 |
| | 11.1 Defi | nitions/Classifications | 38 |
| | 11.1.1 | Evaluation and Documentation of Adverse Events | 39 |
| | 11.1.2 | Evaluation and Documentation of Device Deficiencies | 40 |
| | 11.2 Rep | orting of Adverse Events | 40 |
| | 11.3 Eme | ergency Contact Details for Reporting AEs and Device Deficiencies | 41 |
| 12 | Data R | Review Committees | 41 |
| | 12.1 Clini | ical Events Committee | 41 |
| 13 | . Statist | ical Design and Methods | 42 |
| | 13.1 Ana | lysis Populations | 42 |
| | 13.1.1 | Enrolled Population | 42 |
| | 13.2 Des | cription of Baseline Variables | 42 |
| | 13.3 Prim | nary Analysis | 42 |
| | 13.3.1 | Primary Endpoint | 43 |
| | 13.4 Sam | ple Size | 43 |
| | 13.5 Seco | ondary Endpoints | 43 |
| | 13.6 Add | itional Exploratory Endpoints | 43 |
| | 13.7 Miss | sing Data | 43 |
| 14 | . Ethics | and Regulatory Compliance | 43 |
| 15 | . Study | Administration | 44 |
| | 15.1. | Monitoring | 44 |

| 1/0 | rcian | |
|-----|-------|-----|
| ve | rsion | 4.0 |

#### 

| 15.2. | Data Management | 45 |
|---|---|---|
| 15.3. | Direct Access to Source Data/Documents | 45 |
| 15.4. | Confidentiality | 45 |
| 15.5. | Liability | 46 |
| 15.6. | CIP Amendments | 46 |
| 15.7. | Record Retention | 46 |
| 15.8. | Publication and Use of Information | 46 |
| 15.9. | Suspension or Early Termination | 47 |
| 15.9. | 1 Suspension or Early Termination of the Trial | 47 |
| 15.9.2 | 2 Suspension or Early Termination of a Trial Site | 47 |
| . Othe | r Institutions and Professional Services | 47 |
| . Versi | on History | 47 |
| . Refer | rences | 51 |
| . Appe | ndices | 53 |
| 19.1 Co | nduction Disturbance Management | 53 |
| 19.2 Qu | ality of Life Questionnaires | 57 |
| 19.3 Ech | nocardiography Procedure | 57 |
| 19.3. | 1 Required Exams | 57 |
| 19.3. | 2 General Imaging and Recording Procedures | 58 |
| 19.3. | 3 List of Recommended Images | 58 |
| 19.3. | 4 Data Requirements | 60 |
| 19.3. | 5 Acquisition of Key Variables | 61 |
| 19.3. | 6 Core Lab Analysis | 70 |
| 19.4 Re | commended MSCT Procedures | 72 |
| 19.4. | 1 General requirements | 73 |
| 19.4.2 | 2 ECG-gated contrast enhanced scan of aortic root | 73 |
| 19.4. | Anatomic suitability and valve size selection | 78 |
| 19.5 Res | sheath and Recapture Definitions | 78 |
| | dpoint Definitions | |
| | 15.9.3 . Othe . Versi . Refer . Appe 19.1 Co 19.2 Qu 19.3 Ech 19.3.3 19.3.4 19.3.4 19.3.4 19.4.5 19.4.5 19.4.5 19.5 Res | 15.3. Direct Access to Source Data/Documents |




## 2. Glossary

| Term | Definition |
|-------|--------------------------------|
| 2D | Two Dimensional |
| AE | Adverse Event |
| ADE | Adverse Device Effect |
| AF | Atrial Fibrillation |
| AR | Aortic Regurgitation |
| AS | Aortic Stenosis |
| AVR | Aortic Valve Replacement |
| BAV | Balloon Aortic Valvuloplasty |
| BNP | Brain Natriuretic Peptide |
| CEC | Clinical Events Committee |
| CIP | Clinical Investigation Plan |
| CLS | Compression Loading System |
| СНВ | Complete heart block |
| CRF | Case Report Form |
| CRO | Contract Research Organization |
| СТ | Computed Tomography |
| CVA | Cerebrovascular Accident |
| DCS | Delivery Catheter System |
| ECG | Electrocardiogram |
| e-CRF | Electronic Case Report Form |
| EDC | Electronic Data Capture |




| Term | Definition |
|---------|--------------------------------------------------|
| EF | Ejection Fraction |
| EQ-5D | European Quality of Life – 5 Dimensions |
| HAVB | High Degree Atrioventricular Block |
| ICF | Informed Consent Form |
| IRB/REC | Institutional Review Board/Research Ethics Board |
| IFU | Instructions For Use |
| ІТТ | Intent-to-treat |
| KCCQ | Kansas City Cardiomyopathy Questionnaire |
| LBBB | Left Bundle Branch Block |
| LS | Loading System |
| MI | Myocardial Infarction |
| MRS | Modified Rankin Score |
| MSCT | Multi Slice Computed Tomography |
| NYHA | New York Heart Association |
| TAV | Transcatheter Aortic Valve |
| PCI | Percutaneous Coronary Intervention |
| TAVR | Transcatheter Aortic Valve Replacement |
| QoL | Quality of Life |
| RBBB | Right Bundle Branch Block |
| SAE | Serious Adverse Event |
| SAVR | Surgical Aortic Valve Replacement |
| SOP | Standard Operating Procedures |
| STS | Society of Thoracic Surgeons |




| Term | Definition |
|------|----------------------------------|
| TEE | Transesophageal Echocardiography |

## 3. Synopsis

| Title | Optimize PRO Study |
|---|---|
| Devices | <ul> <li>Medtronic Evolut™ PRO Transcatheter Aortic Valve (TAV)</li> <li>Medtronic Evolut™ PRO+ Transcatheter Aortic Valve (TAV)</li> <li>Medtronic EnVeo™ PRO Delivery Catheter System (DCS) with EnVeo™ InLine Sheath or EnVeo™ R DCS with EnVeo™ InLine Sheath</li> <li>Medtronic Evolut™ PRO+ Delivery Catheter System (DCS)Medtronic EnVeo™ PRO Loading System (LS) or EnVeo™ R LS</li> <li>Medtronic Evolut™ PRO+ Loading System (LS)</li> <li>Guidewires (e.g. Confida, etc)</li> <li>Sheaths (e.g. Confida, etc)</li> </ul> |
| Sponsor | Medtronic Coronary and Structural Heart Clinical Research |
| Co-Principal Investigators | Dr. Steven Yakubov and Dr. Kendra Grubb |
| Primary Objective | The purpose of this study is to collect clinical evidence on valve performance and procedural outcomes associated with an "optimized" TAVR care pathway and using the Evolut™ PRO and Evolut™ PRO+ devices |
| Primary Endpoint | Rate of all-cause mortality or all-stroke at 30 days |
| Secondary Endpoints | <ul> <li>Median days from index procedure to discharge</li> <li>Percentage of subjects with ≥ moderate aortic regurgitation (AR) at discharge.</li> </ul> |
| | <ul> <li>Rate of pacemaker implant for new onset or worsening conduction<br/>disturbance at 30 days</li> </ul> |
| Additional Exploratory | 30-day and 1-year hospital re-admission rates |
| Endpoints | 1-year composite of all-cause mortality or all-stroke |
| Study Design | Post-market, multi-center, prospective, non-randomized |
| Sample Size | Up to 46 sites in the United States and Canada with up to 400 subjects |


| Patient Population | Subjects with severe, symptomatic aortic stenosis (AS) necessitating valve replacement |
|---|---|
| Duration | Total study duration is estimated to be 2 years (time from first subject implanted to one-year follow-up on last subject implanted) |
| Key Inclusion Criteria | <ul> <li>Acceptable candidate for treatment with the Evolut™ PRO or Evolut™ PRO+ system in accordance with the Instructions for Use and local regulations;</li> </ul> |
| | <ul> <li>Subject is symptomatic from his/her aortic valve stenosis, as<br/>demonstrated by New York Heart Association (NYHA) Functional<br/>Class II or greater;</li> </ul> |
| | <ul> <li>Subject and the treating physician agree that the subject will return<br/>for all required post procedure follow-up visits;</li> </ul> |
| | <ul> <li>Anatomically suitable for transfemoral TAVR with the Medtronic<br/>TAVR system;</li> </ul> |
| | Subject meets the legal minimum age to provide Informed Consent based on local regulatory requirements; |
| Key Exclusion Criteria | Contraindicated for treatment with the Evolut™ PRO or Evolut™ PRO+ system in accordance with the Instructions for Use |
| | <ul> <li>Anatomically not suitable for the Evolut<sup>™</sup> PRO or Evolut<sup>™</sup> PRO+<br/>system;</li> </ul> |
| | <ul> <li>Any percutaneous coronary or peripheral interventional procedure<br/>performed within 30 days prior to enrollment;</li> </ul> |
| | Previous aortic valve replacement; |
| | <ul> <li>Reduced ventricular function with left ventricular ejection fraction<br/>(LVEF) &lt; 35% as measured by resting echocardiogram;</li> </ul> |
| | Frailty assessments identify: |
| | <ul> <li>Subject is &lt;80 years of age and three or more of the<br/>following apply; OR subject is ≥ 80 years of age and two<br/>or more of the following apply</li> </ul> |
| | <ul> <li>Wheelchair bound</li> </ul> |
| | <ul> <li>Resides in an institutional care facility (eg.</li> </ul> |
| | nursing home, skilled care center) |
| | Body Mass Index <20kg/m <sup>2</sup> |
| | <ul><li>Grip strength &lt;16kg</li><li>Katz Index score ≤4</li></ul> |
| | ■ Albumin <3.5 g/dL |
| | Bicuspid valve verified; |
| _ | - Dicaspia vaive verifica, |


| Medtronic |
|-----------|


| | <ul> <li>Aortic root angulation (angle between plane of aortic valve annulus<br/>and horizontal plane/vertebrae) &gt; 70°.</li> </ul> |
|---|---|
| | Implanted with pacemaker or ICD; |
| | Prohibitive left ventricular outflow tract calcification; |
| | Estimated life expectancy of less than 12 months due to associated non-cardiac co-morbid conditions; |
| | <ul> <li>Other medical, social, or psychological conditions that in the opinion<br/>of the Investigator precludes the subject from appropriate consent,<br/>adherence to the protocol required follow-up exams;</li> </ul> |
| | <ul> <li>Currently participating in an investigational drug or another device<br/>trial (excluding registries);</li> </ul> |
| | Need for emergency surgery for any reason; |
| | Subject is less than legal age of consent, legally incompetent, or otherwise vulnerable. |
| Study Procedures and | Clinical assessment at baseline, discharge, 30 days, and 1 year |
| Assessments | <ul> <li>Transthoracic echo at baseline, discharge, and 1 year</li> </ul> |
| | Multi-Detector Computed Tomography at baseline |
| | Quality of Life pre and post-procedure, 30 days, and 1 year |
| | 12-lead ECG at pre and post-procedure, 30 days, and 1 year |

### 4. Introduction

## 4.1. Background and Rationale

Transcatheter aortic valve replacement (TAVR) has been shown to be a safe and effective treatment for patients with severe aortic stenosis who are at extreme, high, or intermediate surgical risk<sup>(1-3)</sup>. Since CoreValve™ became commercially approved in the United States by the Food and Drug Administration (FDA) in 2014, the procedure and valve iterations have become increasingly efficient with reducing complications. The Evolut™ PRO and Evolut™ PRO+ valve's outer pericardial wrap was designed to enhance annular sealing to promote a decrease in paravalvular leak<sup>(4)</sup>. There is also a growing shift towards optimizing the TAVR care pathway by protocolizing the pre, peri, and post procedure assessments. This optimization can further increase the efficiency of the procedure and subsequently decrease the length of hospital stay and reduce health care costs<sup>(5,6)</sup>.

This procedural efficiency has not translated to a reduction in permanent pacemaker implantation (PPI) rates. Rates have decreased with newer generation TAVR valves, however, variability continues<sup>(7)</sup>. There is a lack of consensus regarding the management of post-TAVR conduction abnormalities leading towards


Medtronic

heterogenous PPI rates across institutions and potentially unnecessary pacemakers for abnormalities that could have resolved intrinsically over time<sup>(8,9)</sup>. Previous studies indicate most of high degree atrioventricular block (HAVB) and left bundle branch block (LBBB) occur prior to hospital discharge, and early monitoring is key to identifying and managing persistent TAVR-induced conduction abnormalities<sup>(10,11)</sup>.

The objective of this study is to collect outcome data on valve performance and a pre-specified TAVR care pathway. Additionally, this study will protocolize the management of the post-TAVR conduction disturbances and evaluate whether a consistent deployment technique will reduce the variability of new onset conduction disturbances.

This study will collect safety and performance data on guidewires and sheaths that are used during the TAVR procedure.

### 4.2. Purpose

The purpose of this study is to collect clinical evidence on valve performance and procedural outcomes associated with an "optimized" TAVR care pathway and using the Evolut™ PRO and Evolut™ PRO+ devices.

## 5. Objectives and Endpoints

## 5.1. Objectives

#### 5.1.1. Primary Objective

The primary objective of this study is to collect clinical evidence on valve performance and procedural outcomes associated with an "optimized" TAVR care pathway and using the Evolut™ PRO and Evolut™ PRO+ devices.

## 5.2. Endpoints

The following endpoints will be used to evaluate the primary trial objectives:

#### **5.2.1.** Primary Endpoint

The primary endpoint is the rate of all-cause mortality or all-stroke at 30 days.

#### **5.2.2.** Secondary Endpoints

The following are the secondary endpoints:

Median days from index procedure to discharge


Medtronic

- Percentage of subjects with ≥ moderate aortic regurgitation (AR) at discharge
- Rate of pacemaker implant for new onset or worsening conduction disturbance at 30 days

#### 5.2.3. Additional Exploratory Endpoints

The following are additional exploratory endpoints:

- 30-day and 1-year hospital re-admission rates
- 1-year composite of all-cause mortality or all-stroke

#### 5.2.4. Rationale

The basis for the selection of these study endpoints include:

- Clinically relevant outcomes of the Evolut™ PRO and Evolut™ PRO+ devices
- In accordance with objectively measuring the efficacy of an optimized care pathway for TAVR subjects
- Objectively defined and measurable in the majority of subjects
- Consistent with current recommendations for endpoints in TAVR clinical studies<sup>(12)</sup>

### 6. Study Design

This is a post market, multi-center, prospective, non-randomized study. The study methods include the following measures to minimize potential sources of bias:

- An external, independent Clinical Events Committee (CEC) will review and adjudicate, at minimum, all deaths and endpoint related adverse events. Safety endpoint results will be based on CEC adjudications.
- All sites will follow a standardized protocol for acquisition of echocardiographic endpoint data.
- Core labs will evaluate all echocardiograms and ECGs. Echocardiographic trial endpoint results will be based on Core Lab assessments.
- Subjects will be screened to confirm eligibility for enrollment with pre-defined inclusion and exclusion criteria.

#### 6.1. Duration

The enrollment period is estimated to be less than 12 months and subjects will be followed for up to one year post index procedure; therefore, the estimated total duration of the study (first subject enrolled to last subject completing his/her last follow-up exam) is estimated to be less than 2 years.




## 6.2. Trial Organization

### **6.2.1 Participating Sites**

This trial may be conducted at up to 46 sites in the United States and Canada. Investigative sites will meet the following criteria:

- The site will have extensive facility experience with TAVR. Operator 1 and Operator 2 must meet
  the minimum of ≥ 20 TAVR procedures in the prior year, or ≥ 40 TAVR procedures in the prior two
  years.
- The site will have the presence or capacity of establishing an investigative team consisting of the following:
  - Minimum of 2 TAVR implanters with expertise in transcatheter aortic valve replacement as noted above
  - Electrophysiologist
  - o Echocardiographer
  - Trial coordinator

### 6.2.2. Site Principal Investigator

Each site will have a Principal Investigator (PI) who is a TAVR implanter among the Heart Team. The PI will have overall responsibility for the conduct of the study at the site, including protecting the rights, safety, and welfare of the study subjects at their site, the integrity of the trial data generated by their site, and for ensuring the trial is conducted in compliance with the Clinical Investigation Plan and IRB/REB requirements.

#### 6.2.2 Heart Team

Each site will utilize a local Heart Team to assess eligibility of the prospective subject for the trial according to the site's standard process and payer requirements.

At a minimum, the local Heart Team should include the TAVR implanter. The site PI may also serve as a member of the Heart Team.

#### **6.2.3 Publication Committee**

A Publication Committee will provide direction and support in the development of clinical publications. The Publication Committee will consist of steering committee members. The Publication Committee will be responsible to:


Medtronic

- Define the publication plan
- Review, approve, and prioritize publication proposals
- Provide input on the scientific merit and clinical relevance of ancillary publications
- Identify the manuscript/abstract first author(s)/writer(s)/presenter(s)
- Review publications prior to submission

The Committee will be in charge of publication efforts until the completion of the primary endpoint. All publication activities post the primary endpoint will be facilitated by the Medtronic TAVR Global Evidence Committee.

#### 6.2.4 Trial Training

Prior to participating, center activation, or subsequent involvement in study activities, Medtronic will provide training to the investigative team on the trial methods, procedures, and requirements. Training may be conducted via site initiation visits, investigator meetings, and/or other media sessions. Medtronic will maintain documentation of these training sessions. Additionally, Medtronic representative(s) may be present at each site's implant procedures as part of the ongoing procedure support process.

### 7. Product Description

## 7.1 Description of Devices

### 7.1.2 Medtronic Evolut PRO and Evolut™ PRO+ Systems

- The Medtronic Evolut PRO System is a TAVR implantation system comprised of the following 3 components (Medtronic Evolut PRO TAV
- Medtronic EnVeo PRO DCS with EnVeo InLine Sheath or EnVeo R DCS with EnVeo InLine Sheath
- Medtronic EnVeo PRO LS or EnVeo R LS

The system components for the Evolut PRO System are shown in Figure 1 and detailed descriptions provided in Sections 7.1.2.1, 7.1.2.3, 7.1.2.4, 7.1.2.6, and 7.1.2.7.

#### Table 1):

- Medtronic Evolut PRO TAV
- Medtronic EnVeo PRO DCS with EnVeo InLine Sheath or EnVeo R DCS with EnVeo InLine Sheath
- Medtronic EnVeo PRO LS or EnVeo R LS


Medtronic

The system components for the Evolut PRO System are shown in Figure 1 and detailed descriptions provided in Sections 7.1.2.1, 7.1.2.3, 7.1.2.4, 7.1.2.6, and 7.1.2.7.

Table 1. Evolut™ PRO System Components

| Component | US Model Number | Canadian Model<br>Number | Size (mm) | Aortic Annulus<br>Diameter (mm) |
|---|---|---|---|---|
| | EVOLUTPRO-23-US | EVOLUTPRO-23 | 23 | 18 – 20 |
| Medtronic Evolut PRO TAV | EVOLUTPRO-26-US | EVOLUTPRO-26 | 26 | 20 – 23 |
| | EVOLUTPRO-29-US | EVOLUTPRO-29 | 29 | 23 – 26 |
| EnVeo R DCS with EnVeo InLine<br>Sheath (20 Fr/16eFr) | ENVEOR-N-US | ENVEOR-N | Used with 23,<br>26, and 29 mm<br>TAVs | Not applicable |
| EnVeo PRO DCS with EnVeo InLine<br>Sheath (20 Fr/16eFr) | ENVPRO-16-US | ENVPRO-16 | Used with<br>23,26, and 29<br>mm TAVs | Not applicable |
| EnVeo R LS | LS-MDT2-23-US | LS-MDT2-23 | Used with 23<br>mm TAV | Not applicable |
| | LS-MDT2-2629-US | LS-MDT2-2629 | Used with 26<br>and 29 mm TAV | Not applicable |
| EnVeo PRO LS | L-ENVPRO-1623US | L-ENVPRO-1623 | Used with 23<br>mm TAV | Not applicable |
| | L-ENVPRO-16-US | L-ENVPRO-16 | Used with 26<br>and 29 mm TAV | Not applicable |


Medtronic



Figure 1. (A) Evolut PRO TAV; (B) EnVeo PRO DCS and EnVeo InLine Sheath; (C) EnVeo R DCS and EnVeo InLine Sheath (D) EnVeo R LS (E) EnVeo PRO LS

The Medtronic Evolut PRO+ System is a TAVR implantation system comprised of the following 3 components (Table 2):

- Medtronic Evolut PRO+ TAV
- Medtronic Evolut PRO+ DCS
- Medtronic Evolut PRO+ LS


Medtronic

The system components for the Evolut PRO+ System are shown in Figure 2 and detailed descriptions provided in Sections 7.1.2.2, 7.1.2.5, and 7.1.2.8.

Table 2 Evolut™ PRO+ System Components

| Component | US Model Number | Canadian Model<br>Number | Size (mm) | Aortic Annulus<br>Diameter (mm) |
|---|---|---|---|---|
| | EVPROPLUS-23US | EVPROPLUS-23 | 23 | 18 – 20 |
| Medtronic Evolut PRO+ TAV | EVPROPLUS-26US | EVPROPLUS-26 | 26 | 20 – 23 |
| Medtronic Evolut PRO+ TAV | EVPROPLUS-29US | EVPROPLUS-29 | 29 | 23 – 26 |
| | EVPROPLUS-34US | EVPROPLUS-34 | 34 | 26 - 30 |
| | L-EVPROP2329US | D-EVPROP23-29 | Used with 23,<br>26, and 29 mm<br>TAVs | Not applicable |
| Medtronic Evolut PRO+ DCS | L-EVPROP34US | D-EVPROP34 | Used with<br>34mm TAV | Not applicable |
| | D-EVPROP2329US | L-EVPROP23-29 | Used with<br>23,26, and 29<br>mm TAVs | Not applicable |
| Medtronic Evolut PRO+ LS | D-EVPROP34US | L-EVPROP34 | Used with 34<br>mm TAV | Not applicable |


Medtronic



Figure 2. (A) Evolut PRO+ TAV; (B) Evolut PRO+ 23-29mm DCS; (C) Evolut PRO+ 34mm DCS (D) Evolut PRO+ 23-29mm LS (E) Evolut PRO+ 34mm LS

#### 7.1.2.1 Medtronic Evolut PRO Transcatheter Aortic Valve

The Evolut PRO TAV is available in 3 sizes (23, 26, 29 mm), covering an aortic annulus diameter of 18 to 26 mm. For the 26mm and 29mm bioprostheses: If the patient's annulus diameter is within 0.5 mm of the upper or lower bound of the range, use of the larger valve size can be considered, provided additional dimensional criteria as outlined in the CIP are met. The TAV is comprised of 3 leaflets, a sealing skirt, and outer tissue wrap constructed from glutaraldehyde-fixated porcine pericardium, sewn to a compressible and self-expandable Nitinol support frame. The TAV is processed with an anti-mineralization treatment of AOA<sup>TM</sup>, a compound derived from oleic acid, a naturally occurring long-chain fatty acid.


Medtronic

#### 7.1.2.2 Medtronic Evolut PRO+ Transcatheter Aortic Valve

The Medtronic Evolut PRO+ TAV is available in 4 sizes (23, 26, 29, 34mm), covering an aortic annulus diameter of 18 to 30 mm. For the 26mm and 29mm bioprostheses: If the patient's annulus diameter is within 0.5 mm of the upper or lower bound of the range, use of the larger valve size can be considered, provided additional dimensional criteria as outlined in the CIP are met. The TAV is comprised of 3 leaflets, a sealing skirt, and outer tissue wrap constructed from glutaraldehyde-fixated porcine pericardium, sewn to a compressible and self-expandable Nitinol support frame. The TAV is processed with an anti-mineralization treatment of AOA, a compound derived from oleic acid, a naturally occurring long-chain fatty acid.

# 7.1.2.3 Medtronic EnVeo PRO Delivery Catheter System with EnVeo InLine Sheath

The EnVeo PRO DCS facilitates the placement of the TAV within the annulus of the aortic valve. The catheter assembly is flexible and compatible with a 0.035 in (0.889 mm) guidewire. The distal (deployment) end of the system features an atraumatic, radiopaque catheter tip and a capsule that covers and maintains the bioprosthesis in a crimped position. The capsule includes a distal flare to enable full recapture of the bioprosthesis after partial deployment. A stability layer is fixed at the handle and extends down the outside of the catheter shaft. It provides a barrier between the retractable catheter and the introducer sheath and vessel walls, thus enabling the catheter to retract freely. Updates to the system include redesign of the distal tip of the DCS.

The EnVeo InLine Sheath is assembled over the stability layer, which functions as a hemostatic introducer sheath and minimizes the access site size to the capsule diameter. The InLine Sheath for the 23 mm, 26 mm, and 29 mm Evolut PRO system is compatible with a 20 Fr introducer.

The DCS consists of a catheter with an integrated handle to provide the user with accurate and controlled deployment. The handle is on the proximal end of the catheter and is used to load, deploy, recapture, and reposition the bioprosthesis. The handle features a gray front grip used to stabilize the system. The blue actuator turns to deploy the bioprosthesis precisely. Arrows on the actuator indicate the direction of rotation required to deploy the bioprosthesis. If desired, the blue actuator can be turned in the opposite direction to recapture the bioprosthesis if the radiopaque capsule marker band has not yet reached the distal end of the spindle. The blue actuator also features a trigger, which can be engaged to make macro adjustments to the capsule position. A blue hand rest connects to the blue actuator. The end of the handle features a tip-retrieval mechanism, which can be used to withdraw the catheter tip to meet the capsule after the device has been fully deployed.

The catheter packaging contains an integrated loading bath and a removable tray with 3 rinsing bowls for loading and rinsing the bioprosthesis. The integrated loading bath features a mirror, which aids in accurate


Medtronic

placement of the bioprosthesis frame paddles during loading. In addition, the device packaging is swiveled and secured to facilitate the bioprosthesis loading procedure.

# 7.1.2.4 Medtronic EnVeo R Catheter Delivery System with EnVeo InLine Sheath

The EnVeo R catheter delivery system facilitates the placement of the TAV within the annulus of the aortic valve. The catheter assembly is flexible and compatible with a 0.035 in (0.889 mm) guidewire. The distal (deployment) end of the system features an atraumatic, radiopaque catheter tip and a capsule that covers and maintains the bioprosthesis in a crimped position. The capsule includes a distal flare to enable full recapture of the bioprosthesis after partial deployment. A stability layer is fixed at the handle and extends down the outside of the catheter shaft. It provides a barrier between the retractable catheter and the introducer sheath and vessel walls, thus enabling the catheter to retract freely.

The EnVeo InLine Sheath is assembled over the stability layer, which functions as a hemostatic introducer sheath and minimizes the access site size to the capsule diameter. The EnVeo InLine Sheath for the 23 mm, 26 mm, and 29 mm Evolut PRO system is compatible with a 20 Fr introducer.

The delivery catheter system consists of a catheter with an integrated handle to assist the user with accurate and controlled deployment. The handle is on the proximal end of the catheter and is used to load, deploy, recapture, and reposition the bioprosthesis. The handle features a gray front grip used to stabilize the system. The blue actuator turns to deploy the bioprosthesis. Arrows on the actuator indicate the direction of rotation required to deploy the bioprosthesis. If desired, the blue actuator can be turned in the opposite direction to recapture the bioprosthesis if the radiopaque capsule marker band has not yet reached the distal end of the spindle. The blue actuator also features a trigger, which can be engaged to make macro adjustments to the capsule position. A blue hand rest connects to the blue actuator. The end of the handle features a tip-retrieval mechanism, which can be used to withdraw the catheter tip to meet the capsule after the device has been fully deployed.

The catheter packaging contains an integrated loading bath and a removable tray with 3 rinsing bowls for loading and rinsing the bioprosthesis. The integrated loading bath features a mirror, which aids in accurate placement of the bioprosthesis frame paddles during loading. In addition, the device packaging is swiveled and secured to facilitate the bioprosthesis loading procedure.

### 7.1.2.5 Medtronic Evolut PRO+ Delivery System

The Evolut PRO+ catheter facilitates the placement of the bioprosthesis within the annulus of the aortic valve. The catheter assembly is flexible and compatible with a 0.035 in (0.889 mm) guidewire. The distal (deployment) end of the system features an atraumatic, radiopaque catheter tip and a capsule that covers and maintains the bioprosthesis in a crimped position. The capsule includes a distal flare to enable the


Medtronic

bioprosthesis to be partially or fully recaptured after partial deployment. A stability layer is fixed at the handle and extends down the outside of the catheter shaft. It provides a barrier between the retractable catheter and the introducer sheath and vessel walls, thus enabling the catheter to retract freely. A PRO+ InLine sheath is assembled over the stability layer, which functions as a hemostatic introducer sheath and minimizes the access site size to the capsule diameter. The catheter is compatible with an 18 Fr (6.0 mm) introducer sheath for the 23, 26, and 29 mm TAVs and a 22 Fr (7.3 mm) introducer sheath for the 34 mm TAV.

The DCS consists of a catheter with an integrated handle to assist the user with accurate and controlled deployment. The handle is on the proximal end of the catheter and is used to load, deploy, recapture, and reposition the bioprosthesis. The handle features a gray front grip used to stabilize the system. The deployment knob turns to deploy the bioprosthesis. Arrows on the deployment knob indicate the direction of rotation required to deploy the bioprosthesis. If desired, the deployment knob can be turned in the opposite direction to partially or fully recapture the bioprosthesis if the radiopaque capsule marker band has not yet reached the distal end of the radiopaque paddle attachment. Once the radiopaque capsule marker band reaches the distal end of the radiopaque paddle attachment, it is at the point of no recapture. The deployment knob also features a trigger, which can be engaged to make macro adjustments to the capsule position. A blue hand rest connects to the deployment knob. The end of the handle features a tip-retrieval mechanism, which can be used to withdraw the catheter tip to meet the capsule after the device has been fully deployed.

The catheter packaging contains an integrated loading bath and a removable tray with 3 rinsing bowls for loading and rinsing the bioprosthesis. The integrated loading bath features a mirror, which aids in accurate placement of the bioprosthesis frame paddles during loading. In addition to these features, the device packaging is swiveled and secured to facilitate the bioprosthesis loading procedure.

#### 7.1.2.6 Medtronic EnVeo R Loading System

The EnVeo R LS facilitates manual loading of the TAV into the deployment sheath capsule of the DCS by gradually reducing the diameter of the bioprosthesis radially to an appropriate diameter. The manual loading is performed during the procedure prior to implantation. The loading procedure is performed while immersing the LS, the TAV, and the distal end of the DCS in cold sterile saline.

The EnVeo R LS was designed with ribs on the interior surface of the cone designed to decrease the friction between the TAV tissue wrap on the inflow cone during loading. There are two loading system models; one for the 23 mm TAV and another for the 26 mm and 29 mm TAV sizes.

### 7.1.2.7 EnVeo PRO Loading System

Similar to the EnVeo R LS, the EnVeo PRO LS is a system of reduction cones and tubing designed to gradually reduce the diameter of the TAV radially to an optimal diameter to facilitate manual loading of the Evolut PRO TAV into the deployment sheath capsule of the EnVeo R DCS or EnVeo PRO DCS. The EnVeo PRO loading system incorporates minor modifications including a change to the capsule guide tube (CGT) to


Medtronic

include a locking collar, which reduces the ability of the user to load the TAV with a paddle in the incorrect position by preventing movement of the frame paddles once positioned in the spindle pockets. Additionally, manufacturing process changes and a minor design and material change, including the color differentiation between the two loading system sizes, was implemented on the catheter tip guide tube (TGT) components. A third modification is to the inner diameter of the inflow ring designed to allow multiple TAVs to seat securely into the inflow ring.

#### 7.1.2.8 Evolut PRO+ Loading System

The Evolut PRO+ LS compresses the bioprosthesis into the catheter. Note: verify the correct delivery system and loading system are used for the Evolut PRO+ 34 mm valve. This loading system is designed for compatibility with this specific TAV and delivery system.

#### 7.2. Manufacturer

The legal manufacturer and design site of the Evolut PRO and Evolut PRO+ systems is as follows:

Medtronic CoreValve LLC



## 7.3. Intended Population

The study population includes patients with symptomatic native aortic valve stenosis necessitating valve replacement. Patients who undergo an emergency procedure should not be included in this study.

## 7.4. Product Training Requirements

The Evolut PRO and Evolut PRO+ devices will be used within the local approved indication, with exception to any exclusion criteria in this protocol, and obtained by the study sites according to standard hospital procedures for commercial products. Local existing approved procedures for commercial product regarding training, distribution, shipment, storage, and handling will be followed. In the event of a device malfunction or explant, please refer to section 9.5.

## 7.5. Product Labeling, Tracking, and Accountability

Subjects enrolled in this study will be treated using commercial product. Device lot and serial numbers, as applicable, will be collected in the Device Identification CRF. As this is not an investigational trial, Product


Medtronic

Accountability Logs (PALs) will not be utilized. Sites will follow their institutional standard practice for device ordering and replenishment of commercial product for use in this study.

In Canada, only system components licensed for sale by Health Canada will be used in the study.

## 7.6. Product Storage

Sites will follow their institutional standard practice for storing commercial TAVR product.

## 8. Selection of Subjects

## 8.1 Study Population

The study population includes patients with symptomatic native aortic valve stenosis that necessitates valve replacement who meet the criteria for on-label use of the Evolut PRO and Evolut PRO+ system in accordance with Instructions for Use and local regulations.

## 8.2. Subject Enrollment

This study will involve up to 400 subjects (not including roll-in subjects) based on the number of subjects with an attempted TAVR procedure among all active sites. To ensure a widespread distribution of data and to minimize bias in the study results, no site will implant more than 50 subjects without prior authorization from Medtronic. Subjects who exit from the study after implantation will not be replaced.

### 8.2.2. Roll-In Subjects

For all participating centers, the first three subjects implanted will be considered "roll-in" subjects and will not be included in the 400 'as-treated' cohort. The purpose of the roll-in subjects is to provide Investigators the time for training and familiarization with the protocolized implant technique. The Training and Education team will review and provide recommendations for transition of sites from roll-in phase to as treated analysis phase.

Roll-in subjects will complete in-clinical follow-up evaluations as noted in section 9.1.5 Follow-Up Evaluations however the results for the roll-in population will be analyzed separately from the primary analysis cohorts.

#### 8.3. Inclusion Criteria

Prospective subjects must meet all of the following inclusion criteria to be eligible for randomization:




- 1. Acceptable candidate for treatment with the Evolut PRO or Evolut PRO+ system in accordance with the Instructions for Use and local regulations;
- 2. Subject is symptomatic from his/her aortic valve stenosis, as demonstrated by New York Heart Association (NYHA) Functional Class II or greater;
- 3. Subject and the treating physician agree that the subject will return for all required post procedure follow-up visits;
- 4. Anatomically suitable for transfemoral TAVR with the Medtronic TAVR system;
- 5. Subject meets the legal minimum age to provide Informed Consent based on local regulatory requirements.

#### 8.4. Exclusion Criteria

Subjects are not eligible for study participation if they meet ANY of the following exclusion criteria:

- 1. Contraindicated for treatment with the Evolut PRO or Evolut PRO+ system in accordance with the Instructions for Use
- 2. Anatomically not suitable for the Evolut PRO or Evolut PRO+ system;
- 3. Any percutaneous coronary or peripheral interventional procedure performed within 30 days prior to enrollment;
- 4. Reduced ventricular function with left ventricular ejection fraction (LVEF) < 35% as measured by resting echocardiogram;
- 5. Previous aortic valve replacement;
- 6. Frailty assessments identify:
  - Subject is <80 years of age and three or more of the following apply; OR subject is  $\geq$  80 years of age and two or more of the following apply
    - Wheelchair bound
    - Resides in an institutional care facility (e.g. nursing home, skilled care center)
    - Body Mass Index <20kg/m²
    - Grip strength <16kg</li>
    - Katz Index score ≤4
    - Albumin <3.5 g/dL
- 7. Bicuspid valve verified;
- 8. Aortic root angulation (angle between plane of aortic valve annulus and horizontal plane/vertebrae) > 70°.
- 9. Implanted with pacemaker or ICD;




- 10. Prohibitive left ventricular outflow tract calcification;
- 11. Estimated life expectancy of less than 12 months due to associated non-cardiac co-morbid conditions;
- 12. Other medical, social, or psychological conditions that in the opinion of the Investigator precludes the subject from appropriate consent or adherence to the protocol required follow-up exams;
- 13. Currently participating in an investigational drug or another device trial (excluding registries);
- 14. Need for emergency surgery for any reason.
- 15. Subject is less than legal age of consent, legally incompetent, or otherwise vulnerable\*.

\* Notes: Vulnerable subjects include individuals whose willingness to volunteer in a clinical investigation could be unduly influenced by the expectation, whether justified or not, of benefits associated with participation or of retaliatory response from senior members of a hierarchy in case of refusal to participate. EXAMPLE Individuals with lack of or loss of autonomy due to immaturity or through mental disability, persons in nursing homes, children, impoverished persons, subjects in emergency situations, ethnic minority groups, homeless persons, nomads, refugees, and those incapable of giving informed consent. Other vulnerable subjects include, for example, members of a group with a hierarchical structure such as university students, subordinate hospital and laboratory personnel, employees of the sponsor, members of the armed forces, and persons kept in detention. (13)

## 9. Study Procedures

#### 9.1 Schedule of Events

Follow-up protocol required evaluations should be performed at the trial site. The protocol required evaluations for each trial interval are listed as follows and summarized in Table 32.

#### 9.1.1 Screening Procedures

The following assessments must be completed within 12 weeks prior to TAVR index procedure unless otherwise indicated:

- Clinical assessment, history, and concomitant medications
  - Physical examination including height, weight, systolic and diastolic blood pressure, and body surface area.
  - o 5-Meter Gait Speed
  - Grip Strength
- NYHA classification
- MDCT angiogram within 1 year prior to procedure
- TTE within 10 weeks prior to procedure
- Heart Team eligibility assessment


Medtronic

- Laboratory tests glomerular filtration rate (GFR), hemoglobin, international normalized ratio (INR) for subjects on warfarin, and serum creatinine
- Modified Rankin Score conducted by certified site personnel
- Quality of Life Questionnaires
  - o EQ-5D
  - o KCCQ
- STS Risk Score
- Katz Index of Independence in Activities of Daily Living

The Optimize PRO study will include a Confirmation of Qualification process conducted by Medtronic Clinical Analysts and an independent Screening Committee to review the anatomical characteristics of potential subjects identified by the sites for enrollment. Depending on whether a subject's anatomical characteristics meet entry criteria for the study, a recommendation to proceed with treatment or to reevaluate / exit the subject will be provided to the site.

#### 9.1.2 Enrollment

Subjects will be considered enrolled into the study at the time of Informed Consent. Due to the inclusion/exclusion criteria, not all patients enrolled in the study will be treated. All sites will be required to maintain a record of patients screened for the trial meeting general inclusion criteria who have signed the approved Informed Consent document. For subjects that do not meet study criteria, the reason for not continuing in the trial must be documented and recorded in the EDC system.

Pediatric, legally incompetent, or otherwise vulnerable patients are not eligible for the trial. Further, the Medtronic TAVR system will not be used as an emergency treatment.

Subjects must have their TAVR procedure as soon as possible and no later than 30 days post-enrollment.

### 9.1.3 Implant Procedure (TAVR)

Procedural aspects specific to the Medtronic TAVR system should be performed according to the Instructions for Use. Concomitant procedures including percutaneous coronary intervention (PCI) are not permitted to be completed during the index procedure.

The valve deployment will be completed in accordance to the cusp overlap technique via procedural angiogram, and the standard procedures of the implanting physicians and the TAVR clinical pathway protocol requirements noted below. This described TAVR clinical pathway should serve as a guide for accelerated discharge. Institutional clinical TAVR pathways can be followed as long as the modifications are consistent with an accelerated discharge.


Medtronic

#### **Pre-procedure:**

- 12-lead ECG within 48 hours prior to procedure
- Develop "early discharge plan" (including frailty, mental assessment, and home health if required) with multi-disciplinary team along with optimized screening checklist for first and / or second visit leading up to TAVR procedure.
- Standardize room layout team composition in procedure room (planning with multi-disciplinary team).

#### Peri-Procedure:

- No pre-deployment balloon aortic valvuloplasty TAVR procedure unless medically necessary
- General anesthesia should be avoided unless deemed necessary (e.g. for placement of a transesophageal echo), and it is believed that its use will not impede an early discharge
- Percutaneous and transfemoral femoral access only
- No urinary catheter
- Minimize central lines: no Swan-Ganz catheterization or internal jugular vein unless for temporary transvenous pacing

#### **Post Procedure Recovery:**

- Complete 12-lead ECG within 2 hours after the TAVR procedure
  - o If no ECG changes compared to pre-procedure ECG and subject did not have pre-existing RBBB:
    - Remove all remaining lines within 2 hours of TAVR procedure
    - Repeat 12-lead ECG prior to discharge to confirm no new ECG changes
  - Refer to Appendix 19.1 Conduction Disturbance Management if new ECG changes or subject had pre-existing RBBB
- Mobilize within 4 6 hours of TAVR procedure
- Minimal intensive care unit (ICU) utilization: consider post-anesthesia care unit (PACU) in place of ICU or transfer straight to stepdown floor or telemetry unit

#### 9.1.3.1 Procedural Angiogram

Conduct initial deployment in the cusp overlap projection and conduct aortogram to obtain the estimated implant depth at the NCC. At the point of no return move to a 3 cusp coplanar view and then roll LAO (no greater than 25°) until aortic arch is open and parallax at the inflow is minimized. Remove any remaining parallax at inflow by moving cranial/caudal. Conduct pre-release aortogram to obtain estimated depth of implant from this view at the LCC.

Conduct final aortogram from the original RAO cusp overlap projection. All aortograms are to be provided to Medtronic in DICOM format.


## Medtronic

#### 9.1.4 Prior to Discharge

- Physical examination including weight, systolic and diastolic blood pressure, and concomitant medications.
- NYHA classification
- 12-lead ECG (refer to Appendix 19.1 Conduction Disturbance Management for discharge 12-lead ECG requirements for subjects with conduction abnormalities)
- Laboratory tests glomerular filtration rate (GFR), hemoglobin, international normalized ratio (INR) for subjects on warfarin, and serum creatinine
- TTE must be done within 12 hours and 7 days post TAVR
- Adverse event review

#### 9.1.5 Follow-Up Evaluations

All treated subjects will undergo follow-up evaluations at the following time points post procedure. All follow-up periods are defined as the number of days after the date of the index procedure.

#### Day 0 = day of index procedure

- 30 days (30 + 14 days)
- 12 months (365 ± 30 days)

#### 30 Days

- Physical examination including weight, systolic and diastolic blood pressure, and concomitant medications.
- NYHA classification
- 12-lead ECG
- Quality of Life Questionnaires KCCQ and EQ-5D
- In-office pacemaker interrogation for subjects implanted with pacemakers post index TAVR procedure
- Adverse event review

#### 12 Months

- Physical examination including weight, systolic and diastolic blood pressure, and concomitant medications.
- NYHA classification
- 12-lead ECG
- Quality of Life Questionnaires KCCQ and EQ-5D
- TTI
- In-office pacemaker interrogation for subjects implanted with pacemakers post index TAVR procedure
- Adverse event review


Medtronic

#### Other Evaluations

- Creatinine clearance from screening and discharge laboratory tests will be derived by the trial database system using the Cockcroft-Gault equation.
- A Modified Rankin Score assessment should be conducted at 1 and 3 months following any stroke event.

**Table 3. Summary of Visit Schedule and Required Evaluations** 

| | Screening | TAVR<br>Procedure | Discharge | 30 Days | 12<br>Months |
|---|---|---|---|---|---|
| Informed Consent and HIPAA<br>Authorization | х | | | | |
| Clinical Assessment (Physical<br>Assessment and Concomitant<br>Medications) | x | | x | x | x |
| NYHA Classification | Х | | Х | X | X |
| TTE | Х | | X | | X |
| MDCT Angiogram | Х | | | | |
| Procedural Angiogram | | X | | | |
| Laboratory Test | X | | X | | |
| 12-Lead ECG <sup>1</sup> | | Х | X | X | X |
| Modified Rankin Score <sup>2</sup> | Х | | | | |
| Quality of Life Questionnaires <sup>3</sup> | Х | | | X | X |
| STS Risks Assessment | Х | | | | |
| Katz Index of Independence in Activities of Daily Living | х | | | | |
| 5-Meter Gait Speed | X | | | | |
| Grip Strength | Х | | | · | |
| Pacemaker Interrogation <sup>4</sup> | | | | X | X |
| Adverse Event Review | | X | X | X | X |

<sup>&</sup>lt;sup>1</sup> Refer to Appendix 19.1 Conduction Disturbance Management for discharge 12-lead ECG requirements

Throughout this trial, UB-04 summary bills and itemized hospital bills may be collected at select clinical sites in the US. Prior to the collection of billing information, patients will be asked to provide the information and permission to obtain such billing records for the length of their follow-up period. All related data will be kept in a secure and confidential database.

<sup>&</sup>lt;sup>2</sup> A Modified Rankin Score assessment should be conducted at 1 and 3 months following any stroke event.

<sup>&</sup>lt;sup>3</sup> Quality of Life Questionnaires include EQ-5D and KCCQ.

<sup>&</sup>lt;sup>4</sup> In-office pacemaker interrogations at pacemaker implant, 30-days, and 12 months and CareLink™ Transmissions at 3, 6, and 9 months required for subjects implanted with pacemakers post index TAVR procedure.


Medtronic

#### 9.1.6 Additional Evaluations for Pacemaker Implants

Medtronic brand pacemakers are required to be implanted for subjects that require pacemaker implantation post the TAVR index procedure through the duration of their study participation in order to collect device data from pacemakers. Device data will be collected remotely via CareLink™ system at 3, 6, and 9 months post pacemaker implantation and during in-office pacemaker interrogations at pacemaker implant, 30-day, and 12-month follow-up visit.

For subjects that require pacemaker implantation, a final 'Interrogate All' device interrogation file must be obtained and saved in a digital format (Save-to-Media) at pacemaker implant, 30 day, and 12-month follow-up visit. One copy will be stored at the site and another copy will be sent to Medtronic (device data must not be cleared). A device interrogation (final 'Interrogate All')/Save-to-Media (or CareLink™ transmission) should also be completed at the time of study exit (prior to 12 months visit) and in the case of a death (where possible).

#### 9.1.7 Missed Follow-Up Visits

Every effort should be made to ensure subjects return to the clinic for all protocol required follow-ups. If the subject is unable to return for an in-person clinic visit, the Investigator, or designee, should document in the subject record the reason the subject was unable to complete the visit and, if applicable, follow the requirements for deviation reporting as outlined in Deviation Handling section.

The investigator should also make every effort to contact the subject within the visit window to collect the subject's vital status as well as information related to potential adverse events, safety data, and hospitalizations.

#### **9.1.8** Core Labs

Transthoracic echocardiography (TTE), ECGs, explants, and angiogram imaging will be sent to core labs for central assessment. Further details of the echocardiography methods are provided in Appendix 19.3.

#### 9.1.9 Informed Consent

Prior to enrolling in the trial, patients should be fully informed of the details of trial participation as required by applicable regulations, the site's IRB/REB and the Declaration of Helsinki. Informed Consent must be obtained from each patient prior to conducting any protocol-induced activities beyond standard of care, by using the Informed Consent Form (ICF) approved by that site's IRB/REB and by Medtronic, Inc. All Informed Consent Forms, including HIPAA forms and/or short form consents, must be approved by Medtronic, Inc. prior to use. The ICF must be signed and dated by the patient and by the person obtaining the consent. Any additional persons required by the site's IRB/REB to sign the Informed Consent Forms must also comply.


Medtronic

Prior to the patient signing the ICF, the investigator or authorized designee will fully explain to the patient the nature of the research, trial procedures, anticipated benefits, and potential risks of participation in the trial. The investigator or delegate will allow adequate time for the patient to read and review the consent form and to ask questions. Signing the ICF serves to document the written and verbal information that the investigator or authorized delegate provides to the patient, the patient's understanding of the information, and his/her agreement to participate. The investigator or authorized delegate must document in the patient's medical records that the patient was consented and the date on which the consent was obtained. The original signed consent form will be retained in the patient's trial records and a copy of the Informed Consent Form will be provided to the patient.

Patients should give written consent before undergoing any protocol-required testing. However, if any of protocol-required baseline/screening evaluations (e.g. echocardiography, MDCT, coronary arteriography, lab work) have been performed for clinical diagnostic purposes prior to consenting, they can be used as the protocol-required exams, provided they were obtained within the protocol-required time windows and contain the necessary information.

#### 9.2 Revisions in Patient Information and Informed Consent Form

Medtronic will inform the investigators whenever information becomes available that may be relevant to the subject's continued participation in the trial. The revised information will be sent to the investigator for approval by the IRB/REB.

## 9.3 Assessment of Efficacy

The following methods will be used for assessing, recording, and analyzing efficacy. Refer to section 9.1 Schedule of Events for timing of these assessments.

- STS risk score
- Heart team assessment
- MSCT
- TTE
- 12-lead ECG
- NYHA functional classification
- EQ-5D and KCCQ quality of life questionnaires

## 9.4 Assessment of Safety

#### 9.4.1 Adverse Events and Device Deficiencies

Serious adverse events, device deficiencies, and non-serious VARC-2 adverse events will be collected from the time of enrollment until the end of the study or until study exit, whichever comes first.


Medtronic

The safety assessment performed during this study will be based on the relatedness to the TAVR implant procedure and the following devices:

- Commercial Study Devices:
  - Medtronic Evolut™ PRO Transcatheter Aortic Valve (TAV)
  - Medtronic EnVeo™ PRO Delivery Catheter System (DCS) with EnVeo™ InLine Sheath or EnVeo™ R DCS with EnVeo™ InLine Sheath
  - Medtronic EnVeo™ PRO Loading System (LS) or EnVeo™ R LS
  - Medtronic Evolut™ PRO+ Transcatheter Aortic Valve (TAV)
  - o Medtronic Evolut™ PRO+ Delivery Catheter System (DCS)
  - Medtronic Evolut™ PRO+ Loading System (LS)
- Commercial Accessory Devices:
  - Sheath
  - Guidewire

## 9.5 Device Malfunction or Explant

In the event of a device malfunction of the TAV device or its components prior to implant or in the event that a TAV is explanted after implant (due to reintervention or autopsy), the TAV and/or affected components should be returned to Medtronic to the following:

Medtronic, Inc.

Attn: Explant Lab [PE#] 1851 E. Deere Avenue Santa Ana, CA 92705-5720

Additional details surrounding the device return process are contained within the Medtronic explant kit that will be provided upon notification of a device malfunction or explant.

## 9.6 Recording Data

Trial sites will assign a unique ID number to each subject. Records of the subject/subject ID relationship will be maintained by the trial site. Individual subject medical information obtained as a result of this trial will be considered confidential.

This trial will utilize an Oracle Clinical Remote Data Capture (RDC) system that is the property of Medtronic. Required data will be recorded on electronic case report forms (eCRFs) by authorized site personnel as indicated on the Delegation Task List (DTL). Trial personnel delegated for eCRF completion and/or approval per the DTL will be trained on the use of the RDC system and thereafter provided with a user name and password to access the system. The eCRFs must be completed and/or updated to reflect the latest observations on the subjects participating in the trial. The investigator (or approved sub-investigator) will electronically sign the appropriate pages of each eCRF.


Medtronic

Data from the core lab will be entered into the Oracle Clinical RDC system by core lab personnel per their procedures established for the trial. The core lab physician will approve core lab eCRFs.

The Oracle Clinical RDC system maintains an audit trail of entries, changes, and corrections in eCRFs. If a person only authorized to complete eCRFs makes changes to an already signed eCRF, the investigator shall re-approve this eCRF.

All trial-related documents must be retained until notified by Medtronic that retention is no longer required. Medtronic will inform the investigator/institution when these documents are no longer required to be retained.

No trial document or image should be destroyed without prior written agreement between Medtronic and the investigator. Should the investigator wish to assign the trial records to another party or move them to another location, advance written notice must be given to Medtronic.

#### 9.6.1 Source Documents

Entered data must be traceable to source documents. Source documentation is defined as the first time the data appear and may include all clinical records, hospital records, procedural reports, autopsy reports, and any other material that contains original information used for trial data collection or adverse event reporting. Identified discrepancies between source documents and the eCRFs will be resolved through the on-line query resolution process per the Data Management plan.

The eCRFs may not serve as source documents. Source documentation for data elements not routinely captured in medical records (e.g. echocardiography variables, MDCT variables, catheter and procedural data variables, Heart Team assessment, Modified Rankin Score) may vary from center to center. The site may use technical worksheets if identified as source documents.

Source documents must be retained by the participating site for a period of two years after trial conclusion (or longer as required by local law) and made available for monitoring or auditing by the sponsor's representative or representatives of the FDA and other applicable regulatory agencies or IRB/REB.

The Investigator must ensure the availability of source documents from which the information on the eCRFs was derived. Where printouts of electronic medical records are provided as original source documents, or where copies of source documents are retained as original source documents, they should be signed and dated by a member of the investigation site team indicating they are a true reproduction of the original source document.


Medtronic

#### 9.7 Deviation Handling

Protocol deviations will be reported regardless of whether medically justifiable, pre-approved by Medtronic, or taken to protect the subject in an emergency.

A protocol deviation is to be completed for each trial protocol deviation, including, but are not limited to the following:

- Failure to obtain Informed Consent prior to participation
- Incorrect version of the Informed Consent form used
- Failure to obtain IRB/REB approval before the start of the study
- Implanted subject did not meet inclusion/exclusion criteria
- Enrollment of subjects during lapse of IRB/REB approval

Investigators should obtain prior approval from Medtronic before initiating any change or deviation from the CIP, except where necessary to protect the life or physical well-being of a subject in an emergency situation. Such approval shall be documented in writing and maintained in the Investigator Site File. Prior approval is generally not expected in situations where unforeseen circumstances are beyond the investigator's control (e.g. subject did not attend scheduled follow-up visit).

In addition, Investigators are required to adhere to local IRB/REB procedures for reporting deviations.

Medtronic is responsible for analyzing deviations, assessing their significance, and identifying any corrective and/or preventive actions that may be warranted. Repetitive or serious investigator compliance issues may represent a need to initiate a corrective action plan, which may include suspension of enrollment or termination of the investigator's or site's participation in the study.

### 9.8 Subject Withdrawal or Discontinuation

Subjects who discontinue participation prematurely will be included in the analysis of results (as appropriate) and will not be replaced in the enrollment of total trial subjects. If a subject is discontinued from the trial early, the reason for discontinuation should be documented in the subject file and a Study Exit eCRF must be completed. If discontinuation is because of safety concerns or lack of effectiveness, the subject shall be asked to be followed for collection of ongoing safety data outside the clinical investigation.

A subject will not be considered lost to follow-up unless all efforts to obtain compliance are unsuccessful. At a minimum, the effort to obtain follow-up information must include 3 attempts to make contact via telephone and if contact via phone is not successful, a traceable letter from the investigator should be sent to the subject's last known address. Should both telephone and mail efforts to contact the subject be unsuccessful, the subject's primary physician should be contacted. Subjects will then be deemed lost to follow up. All contact efforts to obtain follow-up must be documented in both the subject's medical records and on the trial eCREs.


Medtronic

If a subject discontinues the trial at any time, is withdrawn from the trial early, or completes all protocol required follow-up they should continue to be followed by the implanting site according to their routine clinical practice for aortic valve patients. If, for any reason, this is not possible for a particular subject, or if a subject needs to change their follow-up site at any time point after conclusion of the trial, investigators should refer subjects to a local site with appropriate training and experience in managing patients with implanted aortic valves.

#### 10 Risks and Benefits

#### 10.1 Potential Risks

There are possible risks and side effects connected to the Evolut PRO or Evolut PRO+ TAV implant, but the risks are the same as those for an implant of the Evolut PRO or Evolut PRO+ TAV without participation in this study. Standard risks associated with the Evolut PRO and Evolut PRO+ systems in the study are provided in the Instruction for Use.

Risks and events will be continuously monitored, assessed and documented by the investigator.

#### 10.2 Potential Benefits

Participation in this clinical study will not result in any direct benefit to the patient. Trial subjects implanted with an Evolut PRO or Evolut PRO+ device receive the same medical treatment as if they were not participating in this post-market study. Participation contributes to expansion of the knowledge base with respect to the use of the Evolut PRO and Evolut PRO+ systems in a routine hospital setting.

#### 10.3 Risk-Benefit Rationale

#### 10.3.1 Measures to Mitigate Risks in the Trial Subjects

The following measures will be implemented to minimize risks to the trial subjects:

- Implanting physicians will have considerable experience with TAVR
- Study sites will have significant experience with TAVR
- Patients will undergo thorough imaging assessment during their pre-implant workup
- Patients will be rigorously followed over the course of the study

#### 10.3.2 Alternatives

Presently, therapeutic alternatives for patients with the clinical indication targeted for the Medtronic TAVR System include the following:




- Medical therapy
- Balloon aortic valvuloplasty
- Surgical aortic valve replacement
- TAVR with a non-Medtronic system

#### 10.3.3 Results from the Risk Analysis and Justification for the Study

TAVR is now established as having an acceptable safe profile and is considered an effective treatment option for patients with symptomatic severe aortic stenosis who are at extreme, high, or intermediated risk for surgical aortic valve replacement. The Medtronic CoreValve™ system, the Evolut R system, the Evolut PRO system, and the Evolut PRO+ system (referred jointly as Medtronic TAVR) has been in widespread use since the first generation received CE Mark in 2007, and there is now extensive published experience demonstrating the Medtronic TAVR system is fulfilling its intended role with a favorable risk/benefit ratio. (14-17) Rigorous clinical trials have established its safety and effectiveness, with improved mortality and quality of life compared with medical therapy in extreme, high and intermediate risk patients. (1-4)

There are risks to the subjects for participation in the trial, they are anticipated to be to the same as risks provided in the IFU and guideline compatible therapy outside of the context of the study (i.e. TAVR or SAVR in a commercial, non-study setting).

#### 11 Adverse Events and Device Deficiencies

### 11.1 Definitions/Classifications

Serious adverse events (SAE) and device deficiencies are collected for this study. The definitions to be applied for the purposes of reporting adverse events are provided in Table 4. Non-serious VARC-2 adverse events will be collected for this study and their definitions are provided in Appendix 0.

**Table 4. Adverse Event Definitions for Reporting Requirements** 

| Event Type | Definition |
|---|---|
| Serious Adverse Event<br>(SAE)<br>(ISO14155:2011 3.37) | Adverse event that a) led to death, b) led to a serious deterioration in the health of the subject, resulting in 1) a life-threatening illness or injury, or 2) a permanent impairment of a body structure or a body function, or 3) in-patient or prolonged hospitalization, or 4) medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function, |
| Device Deficiency | c) led to fetal distress, fetal death or a congenital abnormality or birth defect (13) Inadequacy of a medical device with respect to its identify, quality, durability, |
| | reliability, safety or performance. |




| NOTE: device deficiency includes malfunctions, use errors, and inadequate labeling. |
|---|

#### Notes:

- The interpretation of Seriousness will exclude certain interventions considered standard of care during hospitalization (e.g. IV hydration, certain medications delivered intravenously due to available intravenous access or NPO (nothing by mouth) status, and the delivery of electrolytes to maintain electrolyte balance or to address mild electrolyte depletion). Any nonoral medication or fluid delivery used to treat an acute physical decompensation/deterioration episode or to otherwise resuscitate a subject will be considered serious by definition in that it prevents a permanent impairment of a body structure or deterioration of the health of a subject.
- Planned hospitalization for a pre-existing condition, or a procedure required by the CIP, without serious deterioration in health, is not considered a serious adverse event.
- Hospitalization requires admission for at least 24 hours.
- Ballooning as needed during the implant procedure is standard practice and should not be considered a reintervention.

#### 11.1.1 Evaluation and Documentation of Adverse Events

Investigators are required to evaluate and document in the subject's medical records all serious adverse events, non-serious VARC-2 related events, and device deficiencies (per the definitions in Table 4) observed in trial subjects from the time of enrollment until they are exited from the trial. All SAEs should be followed through their resolution.

Documented pre-existing conditions are not considered to be reportable unless there is a change in the nature or severity of the condition and meets definition of a SAE per definition in Table 4 or a non-serious VARC-2 AE in Appendix 19.6. Pre-existing events should be reported as an SAE in the situation where a new treatment has to be started or an existing treatment has to be changed to treat the adverse event and the event is accompanied with signs and symptoms.

Unavoidable events are conditions which do not fulfill the definition of an Adverse Event, meaning those medical occurrences, clinical signs (including toward abnormal laboratory findings), diseases or injuries that are not untoward in nature; specifically, those resulting from the intended injury such as the index TAVR procedure. The events listed in Table 5 are expected for patients undergoing TAVR, and do not need to be reported as AE, unless they occur outside of the stated timeframe, are otherwise considered to be an SAE according to the treating investigator, or are suspected or confirmed to be device-related.

Table 5. Non-Reportable Medical Occurrences Associated with the Index Procedure

| Event | Timeframe (hours)<br>from the Index<br>Procedure |
|---|---|
| Short transient episode of arrhythmia (including ventricular fibrillation) <u>during</u> index procedure | 0 |




| Event | Timeframe (hours)<br>from the Index<br>Procedure |
|---|---|
| Confusion, anxiety and/or disorientation (other than TIA/stroke) starting within 48 hours with or without medical intervention | 120 (5 days) |
| Temporary change in mental status (other than TIA/stroke) not requiring additional medical interventions or new medical assessments (e.g. CT) | 72 |
| Dizziness and/or lightheadedness with or without treatment | 24 |
| Headache with or without treatment | 72 |
| Sleep problems or insomnia with or without treatment | 120 (5 days) |
| Mild dyspnea or cough with or without treatment | 72 |
| Oxygen supply after extubation / "forced breathing therapy" | 48 |
| Diarrhea with or without treatment | 48 |
| Obstipation / Constipation with or without treatment | 72 |
| Anesthesia-related nausea and/or vomiting with or without treatment | 24 |
| Low-grade fever (<101.3°F or <38.5°C) without confirmed infection | 48 |
| Low body temperature | 6 |
| Pain (e.g. back, shoulder) related to laying on the procedure table with or without treatment | 72 |
| Incisional pain (pain at access site) with or without standard treatment and patient not returning to clinic to have additional treatment | No time limit |
| Pain in throat and/or trachea due to intubation | 72 |
| Mild to moderate bruising or ecchymosis | 168 (7 days) |
| Atelectasis / Pleural Effusion not requiring punctuation | 168 (7 days) |
| Edema resulting in weight increase up to 4 kg / 9lbs from baseline | 168 (7 days) |

#### 11.1.2 Evaluation and Documentation of Device Deficiencies

Device deficiency information will be collected throughout the trial and reported to Medtronic. Device deficiencies should be reported on a Device Deficiency eCRF (one for each Device deficiency) or on the AE CRF if the deficiency led to an adverse event (any untoward medical occurrence, unintended disease or injury, or untoward clinical signs).

# 11.2 Reporting of Adverse Events

Investigators are required to report all serious adverse events (SAE) and non-serious VARC-2 adverse events observed in the study subjects from the point of enrollment until completion of follow-up.


Medtronic

The VARC-2 document provides standardization of endpoint definitions for studies evaluating the use of TAVI. This study follows VARC-2 to allow for improved comparability and interpretability of study results. In addition, Investigators are obligated to report adverse events in accordance with the requirements and timeframes per their reviewing IRB/REB and local regulations, if applicable.

The Sponsor is obligated to report adverse events and device deficiencies that occur during this trial to the IRB/REB as per local requirements.

# 11.3 Emergency Contact Details for Reporting AEs and Device Deficiencies

Investigators should contact their Medtronic clinical trial monitor or site manager if they have any questions regarding reportable AEs. Medtronic will provide and maintain a listing of current contact details for each site.

#### 12 Data Review Committees

#### 12.1 Clinical Events Committee

A Clinical Events Committee (CEC) will provide independent medical review and adjudication of adverse event data used in the safety assessment of the device. The CEC will adjudicate, at minimum, all deaths and safety endpoint-related adverse events. The CEC will follow the recommendations of VARC-2 for classifying adverse events that relate to clinical safety endpoints. The analysis of the trial safety data will be based on CEC adjudicated events. Safety endpoint definitions are provided in Appendix 19.6

**Endpoint Definitions.** 

The CEC members will be free from bias towards the trial and will be independent from both the trial and investigators and Medtronic. The committee will consist of at least 3 independent experts (non-Medtronic employed physicians) with expertise relevant to the trial. This may include experience in the areas of:

- Cardiac surgery
- Interventional cardiology
- Neurology
- Electrophysiology




# 13. Statistical Design and Methods

#### 13.1 Analysis Populations

#### 13.1.1 Enrolled Population

Within the enrolled population the following analysis sets are distinguished:

- The as treated (AT) set: The AT set consists of all enrolled subjects with an attempted TAVR implant procedure, defined as when the subject is brought into the procedure room and any of the following have occurred: anesthesia or conscious sedation administered, vascular line placed, TEE placed, or any monitoring line placed. Subjects will be analyzed according to their first attempted procedure. Enrolled subjects that do not receive an attempted TAVR implant are to be exited from the study.
- The implanted set: The implanted set consists of all the AT subjects who are actually implanted with the TAV. Subjects with an attempted implant that do not actually receive a TAV are to be exited from the study following discharge from the index hospitalization.
- **Per protocol set:** The per protocol set consists of all implanted subjects who's index procedure adhere to the TAVR care pathway as described in section 9.1.3 Implant Procedure TAVR (iliofemoral, no concomitant procedures, etc.)
- **Roll-in:** Roll-ins subjects will not be analyzed with the AT, implanted, or per protocol set and will be analyzed separately using descriptive statistics.

The primary analysis for the primary objective and secondary safety and effectiveness objectives will use the as treated set.

# 13.2 Description of Baseline Variables

Baseline demographic and clinical variables will be summarized for the AT, implanted, and per protocol sets. Continuous variables will be summarized as means, medians, standard deviations, interquartile ranges, minima and maxima and categorical variables will be summarized as frequencies and percentages.

### 13.3 Primary Analysis

The study objective and endpoints are descriptive, and no statistical hypothesis testing will be performed. Interim analyses will be conducted after 100 subjects are enrolled in the AT set and followed through 30 days post procedure.

Roll-in subjects will not be included in the primary analysis; however, the data will be summarized separately with descriptive statistics.




#### 13.3.1 Primary Endpoint

The primary endpoint is the rate of all-cause mortality or all-stroke at 30 days. A Kaplan-Meier survival analysis will be performed with results summarized at 30 days and 12 months. This endpoint is descriptive, and no statistical hypothesis test will be performed.

# 13.4 Sample Size

The sample size for the AT population is 400 subjects and up to 46 sites in the US and Canada. The sample size for the roll-in population is up to 138 subjects. Total combined sample size with all analysis populations is up to 538 subjects.

This is not a hypothesis-driven study, therefore the sample size of up to 400 subjects was not determined by statistical sample size methods. With >25% of TAVR patients experiencing new conduction disturbances<sup>10</sup>, 400 patients will provide a sufficient sample (~100 patients) to evaluate the conduction disturbance management pathway.

# 13.5 Secondary Endpoints

The following are the secondary endpoints:

- Median days from index procedure to discharge
- Percentage of subjects with ≥ moderate aortic regurgitation (AR) at discharge
- Rate of pacemaker implant for new onset or worsening conduction disturbance at 30 days

### 13.6 Additional Exploratory Endpoints

The following are additional exploratory endpoints:

- 30-day and 1-year hospital re-admission rates
- 1-year composite of all-cause mortality or all-stroke

# 13.7 Missing Data

Every effort will be undertaken to minimize missing data. However, some missing data is inevitable, and the trial is designed with the expectation that there may be up to 6% of primary data missing at 12 months.

# 14. Ethics and Regulatory Compliance

This study will be conducted in accordance to the Evolut PRO and Evolut PRO+ system commercially approved IFU and therefore is not considered to be a high risk study. An Investigational Device Exemption


Medtronic

(IDE) is not required to be submitted to the FDA and a pre-approval submission is not required to be submitted to Health Canada, if appropriate.

The study will be conducted in accordance with the protocol, GCP, and ethical principles that have their origin in the Declaration of Helsinki. Each site must fulfill all local regulatory requirements prior to enrolling subjects, as applicable.

Participating sites will not be activated nor begin enrolling subjects until the required approval/favorable opinion from the local IRB/REB and regulatory agency has been obtained (as appropriate).

This trial will be publicly registered prior to first enrollment in accordance with the 2007 Food and Drug Administration Amendments Act (FDAAA) and on <a href="http://clinicaltrials.gov">http://clinicaltrials.gov</a> (PL 110-85, Section 810(a)).

Prior to enrolling subjects, each investigation site's IRB/REB will be required to approve the current CIP, the Informed Consent Form, and any other written information to be provided to the subjects. Study sites must also utilize IRB/REB approved Health Insurance Portability and Accountability Act (HIPAA) Authorization, when applicable.

IRB/REB approval of the clinical trial must be received in the form of a letter and provided to Medtronic before commencement of the trial at an investigation site. The approval letter must contain enough information to identify the version or date of the documents approved. IRB/REB roster or letter of compliance needs to be provided to allow verification that the investigator, other center trial staff, and/or Medtronic personnel are not members of the IRB/REB. If they are members of the IRB/REB, written documentation is required stating that he/she did not participate in the approval process. Investigators must inform Medtronic of any change in status of IRB/REB approval once the investigation site has started enrollment. If any action is taken by an IRB/REB with respect to the study, that information will be forwarded to Medtronic by the respective investigator.

# 15. Study Administration

### 15.1. Monitoring

Participating sites will be monitored to ensure compliance with the trial protocol, adherence to applicable regulations, and accuracy of trial data. Monitoring visits will be conducted primarily to ensure the safety and well-being of the subjects is preserved. Sites should provide appropriate access to the source data. Site personnel will complete eCRFs following each subject visit. Trial data submitted will be reviewed against subject charts and other sources containing original records of subject data. Source document verification will occur via a risk-based approach as outlined in the Monitoring Plan.

The progress of the trial will be monitored by:

• On-site review, as deemed appropriate by Medtronic




- Telephone communications between the site personnel (e.g., investigator, trial coordinator) and trial monitors
- Review of eCRFs and the associated clinical records
- Review of regulatory documents

Upon study completion, Site Closeout Visits will be conducted as outlined in the Monitoring Plan

Monitoring and monitoring oversight will be provided by Medtronic



Prior to the first site activation a monitoring plan will be established outlining the above activities, as well as trial materials to be supplied to sites, the process for corrective and preventive actions and Investigator disqualification procedures.

#### 15.2. Data Management

Medtronic will be responsible for the processing and quality control of the data. Data review, database cleaning and issuing and resolving data queries will be done according to Medtronic internal SOPs and the Data Management Plan for this trial. The trial database will be developed and validated per the Data Management Plan for this trial and will employ validation programs (e.g. range and logic checks) on entered data to identify possible data entry errors and to facilitate data validation. The trial database will maintain an audit trail of all changes made to the eCRFs.

# 10.2 Refer to Device Malfunction or Explant

In the event of a device malfunction of the TAV device or its components prior to implant or in the event that a TAV is explanted after implant (due to reintervention or autopsy), the TAV and/or affected components should be returned to Medtronic to the following:

Medtronic, Inc.

Attn: Explant Lab [PE#] 1851 E. Deere Avenue Santa Ana, CA 92705-5720

Additional details surrounding the device return process are contained within the Medtronic explant kit that will be provided upon notification of a device malfunction or explant.

Recording Data section for further information regarding data collection and management procedures.




#### 15.3. Direct Access to Source Data/Documents

Medtronic may conduct audits at participating clinical sites. The purpose of an audit is to verify the performance of the monitoring process and the trial conduct, independent of the personnel directly involved in the trial.

The investigator and/or institution shall permit Medtronic, regulatory bodies, and IRB/REB direct access to source data and documents.

# 15.4. Confidentiality

All information and data sent to parties involved in trial conduct concerning subjects or their participation in this trial will be considered confidential. Trial sites will assign a unique subject ID number (SID) to each subject. Records of the subject/SID relationship will be maintained by the trial site. The SID is to be recorded on all trial documents to link them to the subject's medical records at the site. To maintain confidentiality, the subjects' name or any other personal identifiers should not be recorded on any trial document other than the Informed Consent Form. In the event a subject's name is included for any reason, it will be masked as applicable. In the event of inability to mask the identification (e.g., digital media), it will be handled in a confidential manner by the authorized personnel.

# 15.5. Liability

Medtronic, Inc (including all wholly owned subsidiaries) maintains appropriate clinical trial liability insurance coverage as required under applicable laws and regulations and will comply with applicable law and custom concerning specific insurance coverage. If required, a Clinical Trial Insurance statement/certificate will be provided to the IRB/REB if required.

#### 15.6. CIP Amendments

The investigator may propose any appropriate modification(s) of the CIP. Medtronic will review this proposal and decide whether the modification(s) will be implemented.

Medtronic will submit any significant amendment to the CIP, including a justification for the amendment to the investigators to obtain approval from their IRB/REB. The investigator will only implement the amendment after approval of the IRB/REB, and Medtronic. Administrative amendments to the CIP will be submitted to the IRB/REB for notification. Furthermore, investigators shall sign any approved amendment for agreement.


Medtronic

#### 15.7. Record Retention

At a minimum, the investigator must retain records for at least 2 years or at least two years have elapsed since the formal discontinuation of clinical development of the devices. The investigator should take measures to prevent accidental or early destruction of the trial related materials.

#### 15.8. Publication and Use of Information

Medtronic is committed to the widespread dissemination of all primary and secondary endpoint results. A Publication Plan will be implemented and followed. At the conclusion of the trial, a multisite abstract reporting the primary results will be prepared by the Principal Investigators (in collaboration with others including but not limited to the echo core lab physicians, and the CEC). A multisite publication will similarly be prepared for publication in a reputable scientific journal. The publication of the principal results from any single site experience within the trial is not allowed until both the preparation and publication of the multisite results, and then only with written permission from Medtronic.

Following analysis and presentation of the endpoint results, active participation of all participating investigators, CEC committee members, and core laboratory personnel will be solicited for data analysis and abstract and manuscript preparation. Submission of all abstracts and publications regarding the primary endpoint and secondary endpoints from the trial requires approval by the Principal Investigators after review by the Publications Committee.

A separate Publication Plan will provide detailed information about the publication committee, authorship, publication proposals, and requests for data.

### 15.9. Suspension or Early Termination

### 15.9.1 Suspension or Early Termination of the Trial

If the trial is terminated prematurely or suspended, Medtronic shall promptly inform the clinical investigators of the termination or suspension and the reason(s) for this. The investigator shall then promptly inform the reviewing IRB/REB. Medtronic will, as soon as possible, provide a written statement to the investigators to enable prompt notification of the IRB/REB. If trial enrollment is terminated early, follow-up visits will continue for all enrolled subjects.

# 15.9.2 Suspension or Early Termination of a Trial Site

Medtronic may decide to suspend or prematurely terminate an investigation site (e.g. in case of expiring approval of the reviewing IRB/REB, non-compliance to the CIP, or lack of enrollment). If an investigation site is suspended or prematurely terminated, Medtronic shall promptly inform the investigator(s) of the


Medtronic

termination or suspension and the reason(s) for this. The investigator shall then promptly inform the reviewing IRB/REB.

#### 16. Other Institutions and Professional Services

This study will utilize an Echo Core Lab, ECG Core Lab, a Pathology Core Lab, and a Clinical Events Committee. Information and contact details for each of these parties will be maintained in a separate document and provided to the study sites. A definitive list of all participating parties will be provided in clinical reports. In addition, a list of the names and addresses of participating institutions will maintained and provided to the sites.

#### 17. Version History

| Version | Summary of Changes | Author(s)/Title |
|---|---|---|
| 1.0 | New Document | |
| 2.0 | <ul> <li>Added statements regarding compliance to the TAVR Clinical Pathway and Conduction Disturbance Appendix</li> <li>Updated all references from "TAVI" to "TAVR"</li> <li>Clarified Operator 1 and 2 minimum requirements in Participating Sites section</li> <li>Revised Heart Team composition in Heart Team section</li> <li>Removed Heart Team eligibility assessment in Summary of Visit Schedule and Required Evaluations section</li> <li>Modified the enrollment rate in the Duration and Sample Size sections</li> <li>Removed requirement of subject meeting inclusion / exclusion criteria prior to consent in the Enrollment section</li> <li>Added definition for signs and symptoms of aortic valve disease in Endpoints Definitions section</li> </ul> | |
| 3.0 | <ul> <li>Update secondary endpoint to say Percentage of subjects with ≥ moderate aortic regurgitation (AR) at discharge</li> <li>Subject Enrollment: Added Roll-In Subject Section: <ul> <li>For all participating centers, the first three subjects implanted will be considered "roll-in" subjects. The purpose of the roll-in subjects is to provide Investigators the time for training and familiarization with the protocolized implant technique. The Training and Education team will review</li> </ul> </li> </ul> | |


Medtronic

- recommendations made by the Steering Committee for transition of sites from roll-in phase to as treated analysis phase.
- Roll-in subjects will complete in-clinical follow-up evaluations as noted in section 9.1.5 Follow-Up Evaluations however the results for the roll-in population will be analyzed separately from the primary analysis cohorts.
- Heart Team: added language stating the Heart Team should assess eligibility of the subject according to the site's standard process and payer requirements.
- Trial Organization: updated Publication Committee members to include steering committee members
- Inclusion/Exclusion Criteria: Added exclusion criteria:
  - Subjects with pre-existing permanent pacemaker
  - o Previous aortic valve replacement
  - Exclude subjects with horizontal aorta (aortic angulation > 70 degrees per the IFU)
  - o Prohibitive left ventricular outflow tract calcification
- Implant Procedure: Added statement in introduction of section.
  - In addition, the valve deployment will be completed in accordance to the cusp overlap technique via procedural angiography.
- Follow-Up Evaluations: Added procedural angiography during TAVR procedure in Summary of Visit Schedule and Required Evaluations table.
- Adverse Events and Definitions:
  - Added in AE definition table: "Ballooning as needed during the implant procedure is standard practice and should not be considered a reintervention."
  - Clarified that Serious Adverse Events and Device Deficiencies will be collected from the time of enrollment
- Statistical Design and Methods: Added potential for interim analysis in Primary Analysis.
- Sample size:
  - Updated rationale for sample size
  - Updated sample size to include roll-in subjects
- Conduction Disturbance Management Appendix: Updates to introduction section
  - Removed statement: An occurrence or recurrence of high-degree atrioventricular block (HAVB) or thirddegree atrioventricular block (complete heart block

| Optimize PRO Clinical Investigation Plan | | |
|---|---|---|
| | Version 4.0 | Medtronic |
| | [CHB]) (see definitions of conduction disturbances section) at any time between procedure and discharge is an indication for permanent pacemaker implantation (PPI) (refer to HAVB during the TAVR procedure section). Removed reference to subjects with pre-existing pacemakers. Added statement: Subjects with pre-existing conduction disturbances (eg RBBB) or new conduction disturbances may be discharged prior to the recommended timeframes with continuous ECG monitoring. Pacing wires may be removed prior to recommended timeframe and telemetry may be discontinued prior to the recommended timeframe to allow for early discharge. Revised instruction for the following cohorts: ■ ECG changes (48 hours post op QRS remains > 150 ms, PR remains > 240 ms, or further increase of ≥ 20 ms PR compared to 24-hour post-op ECG) and New LBBB (48 hours post op continuing QRS > 150 ms or PR > 240 ms): Revised instruction: consider EP study to further evaluate if the subject should be implanted with a permanent pacemaker or discharge with continuous ECG monitoring system until 30-day follow-up visit. Endpoint Definitions: Clarified valve thrombus found at autopsy in a subject whose cause of death was not valverelated or found at operation for an unrelated indication should not be reported as valve thrombosis. | |
| | <ul> <li>Added the Evolut PRO+ 23, 26, 29, and 34mm TAVs, DCSs, and<br/>LSs to the commercially available devices able to be used in the<br/>study</li> </ul> | |
| | <ul> <li>Added guidewires and sheaths to the device list in the Synopsis</li> <li>Added requirement to report non-serious VARC-2 adverse</li> </ul> | |
| 4.0 | Added requirement to report non-serious VARC-2 adverse events from the time of enrollment until the completion of follow-up | |
| | Section 8.2.2 Updated to say the Training and Education Committee will provide recommendations for transition of sites from roll-in phase to as treated analysis phase. | |

from roll-in phase to as treated analysis phase.


Medtronic

- Section 9.1.1 Screening Procedures: moved the ECG done at 48 hours pre-procedure from the screening procedures to the preprocedure visit
- Section 9.1.3 Implant procedure (TAVR): updated language under Peri-Procedure to say "General anesthesia should be avoided unless deemed necessary (e.g. for placement of a transesophageal echo), and it is believed that its use will not impede an early discharge
- Added section 9.1.3.1 Procedural Angiogram instructions
- Section 9.1.4 Prior to Discharge: added requirement to collect weight in the physical exam
- Section 9.1.5 Follow-Up Evaluations: removed requirement to collect height
- Section 9.1.5 Follow-Up Evaluations: changed collection of summary bills and itemized hospital bills to 'may be collected' instead of 'will be collected'
- Section 9.1.8 Core Labs: removed statement saying external Holter monitor data will be sent to a core lab
- Added section 9.5 Device Malfunction or Explant
- Section 13.1.1 Enrolled Population Per protocol set: removed 'treated with conscious sedation'
- Section 13.7 Missing Data: removed "The reasons for missing data will be described and evaluated for assessment of possible bias. The distribution of prognostic factors between subjects with data and those without data will be examined to evaluate any potential sources of bias."
- Section 16 Other Institutions and Professional Services: added Pathology Core Lab
- Appendix 19.1 Conduction Disturbance Management: Updates to the pathways based

#### 18. References

- Popma JJ, Adams DH, Reardon MJ et al. Transcatheter aortic valve replacement using a selfexpanding bioprosthesis in patients with severe aortic stenosis at extreme risk for surgery. J Am Coll Cardiol 2014;63:1972-81.
- 2. Adams DH, Popma JJ, Reardon MJ et al. Transcatheter aortic-valve replacement with a self-expanding prosthesis. N Engl J Med 2014;370:1790-8.
- 3. Reardon MJ, Van Mieghem NM, Popma JJ et al. Surgical or Transcatheter Aortic-Valve Replacement in Intermediate-Risk Patients. N Engl J Med 2017;376:1321-1331.


Medtronic

- 4. Forrest JK, Mangi AA, Popma JJ et al. Early Outcomes With the Evolut PRO Repositionable Self-Expanding Transcatheter Aortic Valve With Pericardial Wrap. JACC Cardiovasc Interv 2018;11:160-168
- 5. Lauck SB, Wood DA, Achtem L et al. Risk stratification and clinical pathways to optimize length of stay after transcatheter aortic valve replacement. Can J Cardiol 2014;30:1583-7.
- 6. Lauck SB, Wood DA, Baumbusch J et al. Vancouver Transcatheter Aortic Valve Replacement Clinical Pathway: Minimalist Approach, Standardized Care, and Discharge Criteria to Reduce Length of Stay. Circ Cardiovasc Qual Outcomes 2016;9:312-21.
- 7. van Rosendael PJ, Delgado V, Bax JJ. Pacemaker implantation rate after transcatheter aortic valve implantation with early and new-generation devices: a systematic review. Eur Heart J 2018;39:2003-2013.
- 8. Brignole M, Auricchio A, Baron-Esquivias G et al. 2013 ESC Guidelines on cardiac pacing and cardiac resynchronization therapy: the Task Force on cardiac pacing and resynchronization therapy of the European Society of Cardiology (ESC). Developed in collaboration with the European Heart Rhythm Association (EHRA). Eur Heart J 2013;34:2281-329.
- 9. Sharma E, Chu AF. Predictors of right ventricular pacing and pacemaker dependence in transcatheter aortic valve replacement patients. J Interv Card Electrophysiol 2018;51:77-86.
- 10. Auffret V, Puri R, Urena M et al. Conduction Disturbances After Transcatheter Aortic Valve Replacement: Current Status and Future Perspectives. Circulation 2017;136:1049-1069.
- 11. Urena M, Mok M, Serra V et al. Predictive factors and long-term clinical consequences of persistent left bundle branch block following transcatheter aortic valve implantation with a balloon-expandable valve. J Am Coll Cardiol 2012;60:1743-52.
- 12. Gilard M ea. Registry of Transcatheter Aortic-Valve Implantation in High-Risk Patients. New England Journal of Medicine 2012:1705-1715.
- 13. International Standard ISO 14155:2011(E). Clinical investigation of medical devices for human subjects Good Clinical Practice.
- 14. Webb JG, Wood DA. Current status of transcatheter aortic valve replacement. Journal of the American College of Cardiology 2012;60:483-92.
- 15. Genereux P, Head SJ, Wood DA et al. Transcatheter aortic valve implantation: 10-year anniversary part II: clinical implications. European heart journal 2012;33:2399-402.
- 16. Buellesfeld L, Gerckens U, Schuler G et al. 2-year follow-up of patients undergoing transcatheter aortic valve implantation using a self-expanding valve prosthesis. Journal of the American College of Cardiology 2011;57:1650-7.
- 17. Ussia GP, Barbanti M, Petronio AS et al. Transcatheter aortic valve implantation: 3-year outcomes of self-expanding CoreValve prosthesis. European heart journal 2012;33:969-76.
- 18. Dubois D, Dubois, E.F. A formula to estimate the approximate surface area if height and weight be known. Arch Intern Medicine 1916;17:863-71.
- 19. Baumgartner H, Hung J, Bermejo J et al. Echocardiographic assessment of valve stenosis: EAE/ASE recommendations for clinical practice. European journal of echocardiography: the journal of the Working Group on Echocardiography of the European Society of Cardiology 2009;10:1-25.
- 20. Douglas PS, Waugh RA, Bloomfield G et al. Implementation of echocardiography core laboratory best practices: a case study of the PARTNER I trial. Journal of the American Society of Echocardiography: official publication of the American Society of Echocardiography 2013;26:348-358 e3.


Medtronic

- 21. Clavel MA, Rodes-Cabau J, Dumont E et al. Validation and characterization of transcatheter aortic valve effective orifice area measured by Doppler echocardiography. JACC Cardiovascular imaging 2011;4:1053-62.
- 22. Shames S, Koczo A, Hahn R, Jin Z, Picard MH, Gillam LD. Flow characteristics of the SAPIEN aortic valve: the importance of recognizing in-stent flow acceleration for the echocardiographic assessment of valve function. Journal of the American Society of Echocardiography: official publication of the American Society of Echocardiography 2012;25:603-9.
- 23. Miller FA, Jr. Echocardiography derived valve area of the Edwards SAPIEN aortic valve prosthesis: new methodology is required to comply with old hemodynamic principles. Journal of the American Society of Echocardiography: official publication of the American Society of Echocardiography 2012;25:610-2.
- 24. Genereux P, Head SJ, Hahn R et al. Paravalvular leak after transcatheter aortic valve replacement: the new Achilles' heel? A comprehensive review of the literature. Journal of the American College of Cardiology 2013;61:1125-36.
- 25. Pibarot P, Hahn RT, Weissman NJ, Monaghan MJ. Assessment of paravalvular regurgitation following TAVR: a proposal of unifying grading scheme. JACC Cardiovascular imaging 2015;8:340-60.
- Zoghbi WA, Enriquez-Sarano M, Foster E et al. Recommendations for evaluation of the severity of native valvular regurgitation with two-dimensional and Doppler echocardiography. Journal of the American Society of Echocardiography : official publication of the American Society of Echocardiography 2003;16:777-802.
- 27. Lang RM, Bierig M, Devereux RB et al. Recommendations for chamber quantification: a report from the American Society of Echocardiography's Guidelines and Standards Committee and the Chamber Quantification Writing Group, developed in conjunction with the European Association of Echocardiography, a branch of the European Society of Cardiology. Journal of the American Society of Echocardiography: official publication of the American Society of Echocardiography 2005;18:1440-63.
- 28. Nagueh SF, Appleton CP, Gillebert TC et al. Recommendations for the evaluation of left ventricular diastolic function by echocardiography. Journal of the American Society of Echocardiography: official publication of the American Society of Echocardiography 2009;22:107-33.
- Zamorano JL, Badano LP, Bruce C et al. EAE/ASE recommendations for the use of echocardiography in new transcatheter interventions for valvular heart disease. Journal of the American Society of Echocardiography: official publication of the American Society of Echocardiography 2011;24:937-65.

# 19. Appendices

# 19.1 Conduction Disturbance Management

The following section is intended to provide consistency in the management of subject's conduction disturbance peri and post the TAVR index procedure.


Medtronic

All subjects are required to have 12-lead ECG within the 2 hours following the TAVR procedure and the day of discharge. The 2-hour post procedure ECG, peri-procedural rhythm abnormalities, and pre-existing conduction abnormalities will determine the pathway.

Subjects with pre-existing conduction disturbances (eg RBBB) or new conduction disturbances may be discharged prior to the recommended timeframes with continuous ECG monitoring. Pacing wires may be removed prior to recommended timeframe and telemetry may be discontinued prior to the recommended timeframe to allow for early discharge.

#### No ECG Changes Immediately (2 Hours) Post Procedure:

- No new ECG changes refers specifically to PR and QRS increase < 20 ms on the ≤ 2-hour post-op ECG compared to the pre-procedure ECG.
- Subjects <u>Without Pre-Existing RBBB</u>:
  - Temporary pacing wires can be removed within 2 hours of the TAVR index procedure with continuous telemetry for 24 hours post-op.
  - o If there are no new changes between the ECG done 24 hours post-op compared to the 2-hour post-op ECG done, then the subject is eligible to be discharged 1-day post op.
  - Proceed with pacemaker implantation if there is an occurrence of HAVB/CHB any time during the post-TAVR period.
- Subjects <u>With</u> Pre-Existing RBBB:
  - Maintain temporary pacing until after 24 hours post the TAVR index procedure.
  - If there are no changes between the ≤ 2-hour post-op ECG compared to the 24-hour post-op ECG, then the temporary pacing wire can be removed. Continue telemetry for 1 day and if there continues to be no new ECG changes then the subject is eligible to be discharged 2 days post index procedure
  - If there are ECG changes of at least ≥ 20 ms in the PR or QRS duration compared to the ECG
     2-hour post-op, then refer to instructions for New ECG Changes.
  - Proceed with pacemaker implantation if there is an occurrence of HAVB/CHB any time during the post-TAVR period.

#### ECG Changes (Increase of PR or QRS ≥ 20 ms) in patients with pre-existing conduction disturbance:

- If there are ECG changes of ≥ 20 m/s in the PR or QRS duration on the ≤ 2-hour post op ECG compared to the ECG done pre-procedure, and subjects have pre-existing RBBB, LBBB, IVCD with QRS ≥ 120 ms or 1<sup>st</sup> degree AVB pre-procedure, then temporary pacing must be maintained until 24 hours post the TAVR index procedure.
  - If ECG changes resolve (regression to baseline value, irrespective of QRS/PR interval duration), OR there are no further changes between the ≤ 2-hour post-op ECG compared to the 24-hour post-op ECG and QRS ≤ 150 ms and PR ≤ 240 ms, then the temporary pacing


Medtronic

wire can be removed. Continue telemetry for 1day. If there are no further ECG changes and/or bradyarrythmias, the subject is eligible to be discharged 2 days post index procedure.

- If there are ECG changes of ≥ 20 ms in the PR or QRS duration OR the QRS > 150 ms or PR > 240 ms, then maintain temporary pacing for an additional 24 hours.
  - If ECG changes resolve (regression to baseline value, irrespective of QRS/PR interval duration), OR no further ECG changes and QRS ≤ 150 ms and PR ≤ 240 ms then temporary pacing wire can be removed; continue telemetry for 1 day. If there are no further ECG changes and/or bradyarrythmias, the subject is eligible to be discharged 2 days post index procedure.
  - If there are no further ECG changes, but QRS >150 ms or PR >240 ms OR further ECG changes of ≥20 ms in the PR or QRS duration consider one of the following:
    - Invasive EP study to guide the decision about pacemaker implantation
    - Continuous ECG monitoring until the 30-day follow-up visit.
    - Pacemaker implantation (not in patients with PR >240 ms but QRS <120 ms)</li>
- Proceed with pacemaker implantation if there is an occurrence of HAVB/CHB any time during the post-TAVR period.

#### **New Onset LBBB Post Procedure:**

- Maintain temporary pacing until after 24 hours post the TAVR index procedure.
  - If there are no changes between the ≤ 2-hour post-op ECG compared to the 24-hour postop ECG or the LBBB is resolved, then the temporary pacing wire can be removed and continue telemetry for 1 day:
    - If there continues to be no new ECG changes or arrythmias and the LBBB resolves, then the subject is eligible to be discharged 2 days post index procedure without continuous monitoring.
    - If the LBBB continues and QRS ≤ 150 ms and PR ≤ 240 ms compared to the 24-hour post-op ECG then the subject is eligible to be discharged 2 days post index procedure with a continuous ECG monitoring via a Holter monitor. The subject should maintain the continuous ECG monitoring system until the 30-day follow-up visit.
    - If the LBBB continues and QRS > 150 ms or PR > 240 ms then consider one of the following:
      - Invasive EP study to guide the decision about pacemaker implantation
      - Continuous ECG monitoring until the 30-day follow-up visit
      - Pacemaker implantation




- If there are further ECG changes of at least ≥ 20 ms in the PR or QRS duration between the 2-hour post-op ECG compared to the 24-hour post-op ECG, then maintain temporary pacing for an additional 24 hours.
  - If no further ECG changes compared to 24-hour ECG (PR or QRS increase < 20 ms)or LBBB is resolved, then refer to instruction noted above.
  - If the ECG changes do not resolve and there is further ≥ 20 ms changes in the PR or QRS duration, then consider one of the following:
    - Invasive EP study to guide the decision about pacemaker implantation
    - Continuous ECG monitoring until the 30-day follow-up visit
    - Pacemaker implantation
- Proceed with pacemaker implantation if there is an occurrence of HAVB/CHB any time during the post-TAVR period.

#### HAVB/CHB (transient or persistent) during the TAVR procedure:

- Maintain temporary pacing until after 24 hours post the TAVR index procedure.
  - If the subject continues to experience HAVB/CHB then proceed with implanting a permanent pacemaker.
  - If the HAVB/CHB resolves and there is not recurrent heart block, then the temporary pacing wire can be removed and continue telemetry for 1 day.
    - If the HAVB/CHB reoccurs then proceed with implanting a permanent pacemaker.
    - If the HAVB/CHB does not re-occur and there are no new ECG changes compared to the 24-hour post op ECG, then the subject is eligible to be discharged 2 days post index procedure Refer to instructions above for any changes to the ECG.

#### **Conduction Disturbances Definitions:**

| Conduction Disturbances (infra nodal block) | |
|---|---|
| Right Bundle Branch Block<br>(RBBB) | <ol> <li>QRS duration ≥120 ms</li> <li>rsr', rsR', rSR', or rarely a qR in leads V1 or V2. The R' or r' deflection is usually wider than the initial R wave</li> <li>In a minority of patients, a wide and often notched R wave pattern may be seen in lead V1 and/or V2</li> <li>S wave of greater duration than R wave or &gt;40 ms in leads I and V6</li> <li>Normal R peak time in leads V5 and V6 but peak R wave &gt;50 ms in lead V1</li> </ol> |


| Medtronic |
|-----------|

| Left Bundle Branch Block<br>(LBBB) | <ol> <li>QRS duration ≥120 ms</li> <li>Broad notched or slurred R wave in leads I, aVL, V5, and V6 and an occasional RS pattern in V5 and V6 attributed to displaced transition of QRS complex</li> <li>Absent Q waves in leads I, V5, and V6, but in the lead aVL, a narrow Q wave may be present in the absence of myocardial pathology</li> <li>R peak time &gt;60 ms in leads V5 and V6 but normal in leads V1, V2, and V3, when small initial R waves can be discerned in the precordial leads 5) ST and T waves usually opposite in direction to predominant QRS voltage</li> </ol> |
|---|---|
| Non-specific<br>intraventricular conduction<br>delay (IVCD) with QRS<br>interval ≥120 ms | QRS interval duration ≥120ms where morphology criteria for RBBB or LBBB are not present |

| Atrioventricular Block | |
|---|---|
| First-degree<br>atrioventricular block | P waves associated with 1:1 atrioventricular conduction and a PR interval >20 ms |
| Mobitz I | Mobitz I heart block is characterized by progressive prolongation of the PR interval on consecutive beats followed by a blocked P wave (i.e., a 'dropped' QRS complex) |
| High-degree<br>atrioventricular block<br>(HAVB) | HAVB is defined as any of the following: Second degree AV block type 2 (Mobitz II) in the presence of a QRS ≥120 ms 2:1 AV block in the presence of a QRS ≥120 ms ≥2 consecutive P waves at a constant physiologic rate that do not conduct to the ventricles Transient third degree AV block In the setting of AF, a prolonged pause (> 3 seconds) or a fixed slow (<50 bpm) ventricular response rate |
| Third-degree<br>atrioventricular block<br>(Complete heart block<br>[CHB]) | P waves with a constant rate with dissociated ventricular rhythm (no association between P waves and R waves) or fixed slow ventricular rhythm in the presence of atrial fibrillation |


Medtronic

# 19.2 Quality of Life Questionnaires

Quality of Life Questionnaires used in this trial include:

- Kansas City Cardiomyopathy Questionnaire (KCCQ)
- EuroQol (EQ-5D)

These questionnaires will be provided under separate cover.

## 19.3 Echocardiography Procedure

#### 19.3.1 Required Exams

Transthoracic echocardiography is required at the following intervals:

| Interval | Time Window |
|-----------|--------------------------------------------|
| Screening | Within 12 weeks prior to procedure |
| Discharge | Between 12 hours and 7 days post-procedure |
| 1 year | Day 365 ± 30 days |

#### 19.3.2 General Imaging and Recording Procedures

- A list of recommended images is provided in Section 19.3.3, List of Recommended Images.
- The subject's ID number and exam interval should be annotated on the image.
- A simultaneous ECG with a clearly defined R-wave should be displayed on all clips.
- Digital cine clips should be a minimum of two cardiac cycles in length (preferably three cycles)
- Color Doppler images should be obtained at a minimum frame rate of 20 Hz through optimization of sector width and depth settings.
- Still frames of measured variables (e.g., LVOT diameter, velocities) should be captured. In addition, still
  frames of spectral Doppler tracings without the measurements should be captured to facilitate analysis
  by the Echo Core Lab. Still frames of spectral Doppler tracings should contain a minimum of 3 cardiac
  cycles for subjects in sinus rhythm, and a minimum of 5 cardiac cycles for subjects in atrial fibrillation
  (two sequential frames per variable may be necessary).
- Spectral Doppler waveforms should be recorded at a minimum sweep speed of 50 mm/sec.
- Echocardiograms should be recorded and archived on a DICOM digital format for transmission to the Echo Core Lab.
- Exams will be transmitted to the Echo Core Lab via compact disc (CD-R) or Web-based picture archiving
  and communication system. Details of the image transmission process for each site will be established
  during site initiation process.


Medtronic

- Exams sent to the Echo Core Lab via CD-R should be DICOM files in a true or pure DICOM format.
- The following information should be documented on any CD-R disks sent to the Echo Core Lab:
  - Trial site ID number
  - Subject ID number
  - Exam date
  - Trial interval

#### 19.3.3 List of Recommended Images

#### Parasternal long-axis window

- 1. 2D gray scale standard view (LV in a sagittal section)
- 2. 2D color Doppler for mitral regurgitation (MR)
- 3. 2D color Doppler of aortic (native or prosthetic) regurgitation (AR)
- 4. If AR is present, ZOOM & narrow sector with focus on vena contracta of regurgitant jet
- 5. 2D gray scale ZOOM for LV outflow tract diameter (LVOT)
- 6. Frozen image of measured LVOT diameter
- 7. 2D gray scale; ZOOM at an intercostal space higher for aortic root/aortic prosthesis

#### Parasternal short-axis window

- 8. 2D grayscale LV at mitral valve level
- 9. 2D grayscale LV at papillary muscle level
- 10. Frozen image of measured LV dimensions (without measurements)
- 11. 2D grayscale LV at apical level
- 12. 2D grayscale aortic valve level
- 13. 2D color Doppler of AR: post-implant start scanning from highest position and record first visible AR jet, scan more downwards and look for additional jets confirm origin of AR jets from PLAX

#### Parasternal long-axis view (RV inflow)

- 14. 2D color Doppler of tricuspid regurgitation (TR)
- 15. If TR is present, CW Doppler of TR jet (frozen image without measurements)
- 16. Frozen image of TR jet velocity with measurements

#### **Apical 4-Chamber window**

- 17. 2D grayscale standard view
- 18. 2D color Doppler of MR
- 19. If MR is present, ZOOM & narrow sector
- 20. If MR is present, CW Doppler of MR jet (frozen image)


Medtronic

- 21. 2D color Doppler of TR
- 22. If TR is present, CW Doppler of TR jet (frozen image without measurement)
- 23. Frozen image of TR jet velocity with measurements
- 24. 2D grayscale focussed on LV with decreased depth
- 25. PW Doppler of transmitral flow at mitral valve tips (frozen image)
- 26. Tissue Doppler of the septal mitral annulus (frozen image)
- 27. Tissue Doppler of the lateral mitral annulus (frozen image)

#### Apical long-axis view

- 28. 2D grayscale standard view
- 29. 2D color Doppler of AR
- 30. If AR is present, ZOOM & narrow sector, shift Nyquist 35-40 for PISA measurements
- 31. If AR is present, CW Doppler of AR jet (frozen image without measurement)
- 32. Frozen image of CW Doppler of AR jet (with measurements)
- 33. CW Doppler of aortic/prosthetic valve (frozen image without measurement)
- 34. Frozen image of measured aortic/prosthetic valve velocity
- 35. PW Doppler LVOT (native aortic valve): within 0.5 1 cm below native aortic valve (frozen image without measurements
- 36. PW Doppler LVOT (post –implant) immediately proximal to inflow of stent or valve (frozen image without measurements)
- 37. Frozen image: measured LVOT velocity

#### **Apical 2-Chamber view**

- 38. 2D grayscale standard view
- 39. 2D grayscale focused on LV with decreased depth

#### **Sub-costal Position**

- 40. 2D grayscale; long-axis view
- 41. 2D grayscale; short-axis view
- 42. 2D grayscale: IVC and hepatic vein
- 43. If TR moderate by color Doppler, PW Doppler of hepatic vein (frozen image)
- 44. IF AR mild by color Doppler, PW Doppler from descending aorta (frozen image)

#### **Supra-Sternal Position**

- 45. CW Doppler of aortic valve velocity non-imaging probe (frozen image without measurements)
- 46. Frozen image: measured aortic valve velocity
- 47. If AR mild by color Doppler, PW Doppler from descending aorta (frozen image)

#### **Right Parasternal Position**


Medtronic

- 48. CW Doppler of aortic valve velocity; non-imaging probe (frozen image without measurements)
- 49. Frozen image: measured aortic valve velocity

#### **Results Reporting**

50. Screen prints of all results pages

#### 19.3.4 Data Requirements

Sites should obtain the appropriate images and Doppler recordings in order for the Echo Core Lab to assess and report the variables listed below. Procedures for acquiring key variables are described in Section 19.3.5, Acquisition of Key Variables.

- Height (cm) and Weight (kg)
- Heart rate
- Left ventricular outflow tract (LVOT) diameter in mid systole
- Max aortic/prosthetic valve velocity (V<sub>2</sub>) by CW Doppler
- Aortic valve velocity time integral (VTI) by CW Doppler
- Mean gradient across aortic valve (MGV<sub>2</sub>) by CW Doppler
- LVOT VTI by PW Doppler
- Grade of aortic/prosthetic transvalvular regurgitation (post-implant only)
- Grade of aortic/prosthetic paravalvular regurgitation (post-implant only)
- Grade of prosthetic total (transvalvular plus paravalvular) regurgitation (post-implant only)
- Grade of mitral regurgitation
- · Grade of tricuspid regurgitation
- Max tricuspid regurgitant (TR) jet velocity (if TR is present)
- Left ventricular internal dimension at end diastole
- Left ventricular internal dimension at end systole
- Interventricular septal thickness at end diastole
- Left ventricular posterior wall thickness at end diastole
- Left atrial diameter (anterior-posterior linear dimension) at systole
- Left ventricular ejection fraction by visual estimate
- Grade of diastolic dysfunction (if present)

In addition, the following variables will be derived by the central database from the appropriate measurements reported on the site eCRF.

- Body surface area (Dubois and Dubois)<sup>(18)</sup>
- Peak aortic pressure gradient


Medtronic

- Aortic valve area (AVA)/effective orifice area (EOA) by continuity equation
- Aortic valve area/effective orifice area index (EOAI)
- Doppler Velocity Index
- Estimated right ventricular systolic pressure (RVSP)

Derived variables will be displayed on the eCRF upon entry of the appropriate raw measurements. The preimplant qualifying AVA must be based on the site reported variables for LVOT diameter, LVOT VTI, aortic valve VTI, height, and weight.

#### 19.3.5 Acquisition of Key Variables

#### 19.3.5.1 LVOT Diameter

Pre-implant LVOT diameter is measured from the inner edge to inner edge of the septal endocardium, and the anterior mitral leaflet in mid-systole (Figure A and B). (19,20). Following implantation of the TAV, LVOT diameter is measured from the parasternal long-axis view, immediately proximal to the inflow aspect of the stent, and in mid systole ( C and D). (19-21) Post-surgical valve implantation, LVOT diameter is measured from the junction of the anterior sewing ring and the ventricular septum to the junction of the sewing ring and the anterior mitral valve leaflet (Figure E and F). (19)


Medtronic



Figure 2 (A) and (B) Examples of measurement of pre-implant LVOT diameter. LVOT diameter is measured from the white-black interface of the septal endocardium to the anterior mitral leaflet, parallel to the aortic valve plane, approximately 0.5 cm below the level of the aortic annulus, and in mid systole (C) and (D) Post TAV implantation, LVOT diameter measurement is from outer edge to outer edge of the inflow aspect of the stent (E) and (F) post surgical valve implantation, LVOT diameter is measured from the junction of the anterior sewing ring and the ventricular septum to the junction of the sewing ring and the anterior mitral valve leaflet.

#### 19.3.5.2 LVOT Velocity

LVOT velocity is recorded with PW Doppler from the apical position, in either the apical long-axis view or in the anteriorly angulated four-chamber view (or "5-chamber view"). For pre-implant exams, the PW sample


Medtronic

volume should be positioned just proximal to the aortic valve, with care to avoid the zone of pre-valve acceleration (usually 0.5 to 1.0 cm proximal to the cusps, Figure ). (19)

Post TAV implantation, the sample volume should be placed proximal to the inflow aspect of the stent.<sup>(22)</sup> Full-screen imaging of the TAV should be used to verify positioning of the sample volume below the stent before switching to spectral Doppler mode (****C and D).<sup>(22,23)</sup>

The LVOT VTI is measured by tracing the modal velocity (middle of the dense signal) for use in the continuity equation. (19)



**Figure 3 (A)** Sample volume placement just proximal to zone of pre-valve acceleration (illustration by Mayo Clinic, used with permission) **(B)** Optimal LVOT velocity signal showing a smooth spectral Doppler recording with a narrow velocity range at each time point **(C)** Illustration showing correct sample volume placement just proximal to inflow of TAV stent **(D)** Full-screen imaging of stent to ensure positioning of sample volume below the TAV stent.


Medtronic

#### 19.3.5.3 Aortic Valve Velocities

Aortic valve velocity should be interrogated with CW Doppler from a minimum of 2 transducer positions (apical and either a parasternal or suprasternal position). The position that provides the highest velocity is used for measurements. A smooth velocity curve with a clear outer edge and maximal velocity should be recorded. The maximal velocity is measured at the outer edge of the dark signal; fine linear signals at the peak should not be included in measurements. The outer edge of the dark "envelope" of the velocity curve is traced to provide both the VTI for the continuity equation and the mean gradient (Figure ). (19)



**Figure 4 (A)** Aortic valve velocities interrogated from multiple transducer positions (*illustration by Mayo Clinic, used with permission*) **(B)** CW Doppler of severe aortic stenosis showing tracing of the velocity curve from mean gradient and VTI, and measurement of max velocity.

#### 19.3.5.4 Assessment of Prosthetic Aortic Regurgitation

An integrated exam approach using color flow, pulsed-wave (PW), and continuous-wave (CW) Doppler is used to assess the severity of transvalvular and paravalvular aortic regurgitation (AR). Color flow Doppler imaging should be performed from the parasternal long and short-axis views, and the apical long-axis and/or 5-chamber views. In the short axis view, color imaging should be performed at multiple levels (from level of the leaflets to below the skirt and frame to assess paravalvular regurgitation, and at the coaptation point of the leaflets for transvalvular (central) regurgitation. (24,25)

If AR is seen by color Doppler, a CW Doppler recording of the regurgitant signal should be obtained for measurement of pressure half-time and assessment of jet density. If the degree of AR by color Doppler appears more than mild by visual estimate, the velocity in the proximal descending aorta should be recorded with PW Doppler.


Medtronic

The degree of transvalvular, paravalvular, and total (transvalvular plus paravalvular) AR will be graded as none, trace, mild, mild to moderate, moderate, moderate to severe, and severe based on the synthesis of the Doppler parameters shown in Table 6. (25) The category of "trace" should be used in cases where regurgitation is barely detectable by color Doppler. Regurgitant signals observed to originate within the stent will be considered transvalvular, and regurgitant signals observed to originate outside the stent will be considered paravalvular.




# Table 6.Parameters for evaluation of the severity of aortic regurgitation

| 3-class Grading Scheme | Trace | Mild | Mild | Moderate | Moderate | Severe |
|---|---|---|---|---|---|---|
| Unifying 5-Class Grading Scheme | Trace | Mild | Mild-to-<br>Moderate | Moderate | Moderate-to-<br>severe | Severe |
| Doppler parameters (qualitative or semiquantitative) | | | | | | |
| Jet Features | | | | | | |
| Extensive/wide jet origin | Absent | Absent | Absent | Present | Present | Present |
| Multiple jets | Possible | Possible | Often present | Often present | Usually present | Usually present |
| Jet path visible along stent | Absent | Absent | Possible | Often present | Usually present | Usually present |
| Proximal flow convergence visible | Absent | Absent | Absent | Possible | Often present | Often<br>present |
| Vena contracta width (mm) | <2 | <2 | 2-4 | 4-5 | 5-6 | >6 |
| Vena contracta area (mm²) | <5 | 5-10 | 10-20 | 20-30 | 30-40 | >40 |
| Jet width at origin (% LVOT diameter) | Narrow (<5) | Narrow (5-<br>15) | Intermediate (15-30) | Intermediate (30-45) | Large (45-60) | Large (>60) |
| Jet density: CW Doppler | Incomplete or faint | Incomplete or faint | Variable | Dense | Dense | Dense |
| Pressure half-time (ms): CW<br>Doppler | Slow (>500) | Slow (>500) | Slow (>500) | Variable (200-500) | Variable (200-<br>500) | Steep (<200) |
| Diastolic flow reversal in descending aorta | Absent | Absent or brief early diastolic | Intermediate | Intermediate | Holodiastolic<br>(end-diast. Vel.<br>>20 cm/s) | Holodiastolic<br>(end-diast. |


Medtronic

| | | | | | | Vel. >25<br>cm/s) |
|---|---|---|---|---|---|---|
| Circumferential extent of PVR (%) | <10 | <10 | 10-20 | 20-30 | >30 | >30 |
| Doppler parameters (quantitative) | | | | | | |
| Regurgitant volume (ml/beat) | <15 | <15 | 15-30 | 30-45 | 45-60 | >60 |
| Regurgitant fraction (%) | <15 | <15 | 5-10 | 10-20 | 20-30 | >30 |
| Effective regurgitant orifice area (mm²) | <5 | <5 | 5-10 | 10-20 | 20-30 | >30 |




#### 19.3.5.5 Assessment of Mitral Regurgitation

Color flow Doppler imaging of the left atrium should be performed from the parasternal long-axis view, and from the apical 4, 2, and long axis views.

Mitral regurgitant (MR) jets should be recorded with CW Doppler using a velocity scale that allows assessment of the density, shape, duration, and peak velocity of the MR jet. If the severity appears moderate or greater by visual assessment, pulmonary vein velocities should be recorded with PW Doppler to assess for the presence of systolic flow reversal. Grading of the severity of mitral regurgitation should be integrative using the parameters in Table 7.<sup>(26)</sup>

Table 7. Parameters for evaluation of the severity of mitral regurgitation

| Parameter | Mild | Moderate | Severe |
|---|---|---|---|
| Color flow jet area | Small, central jet<br>(usually <4 cm <sup>2</sup> or<br><20% of LA area) | Variable | Large central jet (usually >10 cm² or >40% of LA area), or variable wall-impinging jet swirling in the LA |
| Jet density (CW) | Incomplete or faint | Dense | Dense |
| Jet contour (CW) | Parabolic | Usually parabolic | Early peaking, triangular |
| Pulmonary vein flow | Systolic dominance | Systolic blunting | Systolic flow reversal |

#### 19.3.5.6 Assessment of Tricuspid Regurgitation

Color flow imaging of the right atrium should be performed from the apical 4-chamber view, the parasternal long-axis view of the RVOT, and the parasternal short-axis view at the level of the aortic valve.

Tricuspid regurgitant (TR) jets should be recorded with CW Doppler using a velocity scale that allows assessment of the density, shape, duration, and peak velocity of the TR jet. If the severity appears moderate or greater by visual assessment, hepatic vein velocities should be recorded with PW Doppler to assess for the presence of systolic flow reversal. Grading of the severity of tricuspid regurgitation should be integrative using the parameters in Table 8.<sup>(26)</sup>

Table 8. Parameters for evaluation of the severity of tricuspid regurgitation

| Parameter | Mild | Moderate | Severe |
|----------------|-------------|-----------------------|--------|
| Jet area (cm²) | <5 | 5 – 10 | >10 |
| VC width (cm) | Not defined | Not defined, but <0.7 | ≥0.7 |




| PISA Radius (cm) | ≤0.5 | 0.6 – 0.9 | >0.9 |
|---|---|---|---|
| Jet density & contour | Soft & parabolic | Dense, variable contour | Dense, triangular, with early peaking |
| Hepatic vein flow | Systolic dominance | Systolic blunting | Systolic flow reversal |

#### 19.3.5.7 Assessment of Left Ventricular Function and Left Atrial Size

Dimensions of the left ventricle and left atrium should be obtained by either 2-D linear measurements or using 2-D guided m-mode from either the parasternal long or short axis views (Figure ). Left ventricular chamber dimensions, septal thickness, and posterior wall thickness are measured using the American Society of Echocardiography (ASE) measurement convention<sup>(27)</sup> (blood-tissue interface). In addition, standard 2-D views of the left ventricle should be obtained from parasternal and apical transducer positions for visual estimation and quantitative assessment of left ventricular ejection fraction using the modified Simpson's rule, and for assessment of regional wall motion.



Figure 5. Measurements of the left ventricle (A) and left atrium (B) using 2-D guided m-mode.

#### 19.3.5.8 Assessment of Left Ventricular Diastolic Function

A spectral Doppler recording of mitral inflow should be obtained with PW Doppler in the apical 4-chamber view, using a 1 to 3 mm sample volume placed between the mitral leaflet tips during diastole (Figure ). The spectral gain and wall filter settings should be optimized to clearly display the onset and cessation of left ventricular inflow. The following variables should be measured:

- Mitral inflow "A" velocity
- Mitral inflow "E" velocity
- Mitral inflow E-wave deceleration time








Figure 6. Positioning of the sample volume for recording of mitral inflow velocities.

Mitral annular velocities should be obtained from the lateral and septal aspects of the mitral annulus using PW tissue Doppler (DTI) performed in the apical 4-chamber view. The sample volume should be positioned at or 1 cm within the septal and lateral insertion sites of the mitral leaflets and adjusted as necessary (usually 5 to 10 mm) to cover the longitudinal excursion of the mitral annulus in both systole and diastole. Minimal angulation (<20 degrees) should be present between the ultrasound beam and the plane of cardiac motion. The following variables should be measured:

- Mitral annular tissue Doppler systolic velocity (septal and lateral)
- Mitral annular tissue Doppler early diastolic velocity (septal and lateral)
- Mitral annular tissue Doppler late diastolic velocity (septal and lateral)

#### 19.3.6 Core Lab Analysis

Protocol-required echocardiograms will be sent to the Echo Core lab for assessment: the data generated by the Echo Core Lab will be the primary data used for analysis and reporting. Received echocardiograms will be logged in and analyzed by the Echo Core Lab according to their procedures determined for this trial.

The Echo Core Lab will report the following variables:

- Heart rate
- Left ventricular outflow tract (LVOT) diameter in mid systole
- Max aortic/prosthetic valve velocity (V<sub>2</sub>) by CW Doppler




- Aortic valve velocity time integral (VTI) by CW Doppler
- Mean gradient across aortic valve (MGV<sub>2</sub>) by CW Doppler
- LVOT VTI by PW Doppler
- Grade of aortic/prosthetic transvalvular regurgitation (post-implant only)
- Grade of aortic/prosthetic paravalvular regurgitation (post-implant only)
- Grade of prosthetic total (transvalvular plus paravalvular) regurgitation (post-implant only)
- · Grade of mitral regurgitation
- Grade of tricuspid regurgitation
- Max tricuspid regurgitant (TR) jet velocity (if TR is present)
- Left ventricular internal dimension at end diastole
- Left ventricular internal dimension at end systole
- Interventricular septal thickness at end diastole
- Left ventricular posterior wall thickness at end diastole
- Left atrial diameter (anterior-posterior linear dimension) at systole
- Left ventricular ejection fraction by visual estimate
- Grade of diastolic dysfunction (if present)
  - Diastolic function should be categorized as normal, mild dysfunction (impaired relaxation pattern), moderate dysfunction (pseudonormal filling), or severe dysfunction (restrictive filling) per the 2009 American Society of Echocardiography recommendations. (28)

Qualitative grading of valvular regurgitation will be performed using the criteria described in Sections 19.3.5.4 through 19.3.4.8. For reporting the degree of prosthetic regurgitation, the grading classes may be collapsed according to the 3-class grading scheme recommended by the American Society or Echocardiography (ASE)-European Association of Cardiovascular Imaging Guidelines. (26,29)

In addition, the following variables will be derived by the central database from the appropriate measurements reported by the Echo Core Lab:

- Peak Pressure Gradient (Peak  $\Delta$  P) Across the Aortic Valve in mmHg Peak  $\Delta$  P = 4 x (V<sub>2</sub><sup>2</sup>)
  - Where: V<sub>2</sub> is the peak velocity across the prosthesis in m/sec
- Aortic Valve Area (AVA) in cm<sup>2</sup> AVA = LVOT diameter in cm<sup>2</sup> x 0.785 x (VTI<sub>V1</sub>/VTI<sub>V2</sub>) Where: VTI<sub>V1</sub> is the velocity time integral of the left ventricular outflow tract in cm, and VTI<sub>V2</sub> is the velocity time integral of the native aortic valve in cm
- Aortic Valve Area Index (AVAI) in cm<sup>2</sup>/m<sup>2</sup>


Medtronic

AVAI = AVA/BSA\*

Where: AVA is the native aortic valve area in cm<sup>2</sup>, and BSA\* is the body surface area in m<sup>21</sup>

• Effective Orifice Area (EOA) in cm<sup>2</sup>

EOA = LVOT diameter<sup>2</sup> x 0.785 x (VTI<sub>V1</sub>/VTI<sub>V2</sub>)

Where:  $VTI_{V1}$  is the velocity time integral of the left ventricular outflow tract in cm, and  $VTI_{V2}$  is the velocity time integral of the aortic prosthesis in cm

Effective Orifice Area Index (EOAI) in cm<sup>2</sup>/m<sup>2</sup>

EOAI = EOA/BSA\*

Where: EOA is the effective orifice area in cm<sup>2</sup>, and BSA\* is the body surface area in m<sup>2</sup>

• Doppler Velocity Index (DVI)

DVI= VTI<sub>V1</sub>/VTI<sub>V2</sub>

Where:  $VTI_{V1}$  is the velocity time integral of the left ventricular outflow tract in cm, and  $VTI_{V2}$  is the time velocity integral of the prosthetic aortic valve in cm

• Left Ventricular Mass (LVM) in grams

 $LVM = 0.83 \times [(LVIDD + LVPW + IVS)3 - (LVIDD)3] + 0.6$ 

Where: LVIDD is the left ventricular internal dimension at end diastole in cm, LVPW is the left ventricular posterior wall thickness at end diastole in cm, and IVS is the interventricular wall thickness at end diastole in cm.

Left Ventricular Mass Index (LVMI) in g/m<sup>2</sup> body surface area

LVMI = LVM/BSA\*

Where: LVM is left ventricular mass in g, and BSA\* is body surface area in m<sup>2</sup>

• Estimated Right Ventricular Systolic Pressure (RVSP) in mmHg

 $RVSP = (4 \times MVTR jet^2) + 10$ 

Where: MV TR jet is the max velocity of the tricuspid regurgitant jet, and 10 = the assumed mean right atrial pressure in mmHg

Body Surface Area\* (BSA) in m<sup>2</sup>

BSA = 0.007184 v (height in cm<sup>0.725</sup> v weight

BSA = 0.007184 x (height in cm<sup>0.725</sup> x weight in kg<sup>0.425</sup>)

### 19.4 Recommended MSCT Procedures

Multi-slice Computed Tomography (Cardiac MSCT) is used to evaluate aortic valve anatomy, determine aortic root dimensions for device sizing, and to evaluate peripheral vessel dimensions and anatomy. The

-

<sup>\*</sup> BSA derived from height and weight reported on the site eCRF

<sup>\*</sup> BSA derived from height and weight reported on the site eCRF




following sections are intended as recommended guidelines for acquiring the images for assessing anatomical suitability for implantation.

### 19.4.1 General requirements

- Multi-detector CT scanner (64-slice minimum) with ECG-gating capability.
- ECG-gated contrast enhanced aortic root (slice thickness of ≤ 1.0 mm)
- Temporal resolution should be optimized to reduce motion artifact.
- Spatial resolution should be as high as possible (goal is smallest isotropic voxel size)

### 19.4.2 ECG-gated contrast enhanced scan of aortic root

Retrospective ECG-gated scans are recommended, which allows for reconstruction in various phases of the cardiac cycle and optimal evaluation of anatomic dimensions and valve morphology. Recommended scan parameters are listed in Table 9.

Prospective ECG-gated sequential scans (step-and-shoot) and high-pitch spiral scans with ECG-gating (flash spiral) are also acceptable. The following parameters are important to the optimum scan:

- Detector collimation 0.4-0.625 mm.
- Slice thickness ≤ 1.0 mm.
- The recommended coverage area is from superior to the aortic arch to inferior to the cardiac apex. The minimum required coverage area is from 50 mm above the aortic annulus to 10 mm below the aortic annulus.
- The recommended slice overlap is 0.4 mm (will result in isotropic voxels with a 20 cm field of view).

### 19.4.2.1 Post-processing

- Retrospective ECG-gated scans
  - Verify heart rate ECG triggers are at consistent place in cardiac cycle, edit if necessary.
     Additional editing/removal of arrhythmias may be performed.
  - Reconstruct at multiple phases (10 increments of 10%), with < 1.0 mm slice thickness. If the system has the capability, also reconstruct a "best systolic" and "best diastolic" phase.
- Prospective ECG-gated scans (including flash spiral)
  - Reconstruct with medium soft kernel and slice thickness ≤ 1.0 mm (slice overlap of 0.4 mm recommended)

#### Table 9. Recommended scan parameters

| Parameter | Recommendation |
|---|---|
| IV injection with iodine | |
| contrast | 80-100 (320mg/ml or higher), modify per patient as appropriate |




| Injection rate | 4-6 mL/sec |
|---|---|
| Bolus tracking, delay | Delay time calculated using protocol for current scanner (bolus tracking or similar) with peak of contrast concentration in the ascending aorta during acquisition. |
| ECG-gating | Retrospective |
| Scan direction | Cranial-caudal |
| Scan coverage | From above the aortic arch to past the cardiac apex |
| Detector collimation | 0.4 – 0.625 mm |
| Pitch | 0.2–0.43 adapted to the heart rate |
| Dose modulation | Modulation and full current between 30 and 80% of the cardiac cycle |
| Slice thickness | 0.8 mm |
| Slice overlap | 0.4 mm |
| Reconstruction kernel | Medium Smooth |
| | Retrospective ECG gating reconstruction algorithm that minimizes motion artifact. |
| Post-processing | Reconstruct at multiple phases (10 minimum). Reconstructed slice thickness ≤ 0.8 mm. |

### 19.4.2.2 Required aortic root measurements

The following measurements of the aortic root are obtained for assessing anatomical suitability:

- Aortic valve annulus perimeter (measured at systole if retrospective gating is used)
- Mean sinus of Valsalva diameter (measured at diastole)
- Mean sinus of Valsalva heights (measured at diastole)

#### Reformatting of Images (21)

- Site image cross-hairs on a ortic root in all windows where it is visible. Lock cross-hairs so they remain orthogonal for all steps.
- In the coronal window, rotate cross-hairs (horizontal line) counter-clockwise to align with virtual basal plane, (Figure ., upper left panel).
- In the sagittal window, the horizontal line is rotated clockwise or counter-clockwise to align with virtual basal plane (Figure , lower left panel).
- On the newly defined double-oblique axial image, scroll up and down through the aortic
  root until the most caudal attachment points of the three native leaflets come into view
  (indicated by arrowheads in Figure 8). If one of the leaflets comes into view at a more
  cranial or caudal slice, adjust the coronal or sagittal cross-hairs until all three leaflets come
  into view on the same axial slice.
- For confirmation of the correct aortic annulus plane, scroll through the double oblique axial
  images starting in the mid sinus and ending at the level of the aortic annulus. The sinuses
  should appear to be relatively the same size at the level of the mid-sinus and the leaflets
  should all disappear equally at the level of the annulus.






Figure 7: Example images in original orientation (axial, coronal, and sagittal). Red curved arrow and line indicate adjustment of coronal and sagittal planes to align with aortic basal annulus.






Figure 8. Example images of reformatted oblique coronal (upper left), oblique sagittal (lower left), double oblique axial (upper right), and 3D reconstruction (lower right). Yellow arrowheads indicate most caudal attachment of three leaflets of the aortic valve).

#### **Aortic annulus measurements**

- Choose the cleanest systolic images for the aortic annulus measurements, either automatically (e.g., best systolic) or by manually identifying. Measurement on a diastolic image is also acceptable.
- Aortic annulus measurements should be completed on the properly reformatted doubleoblique axial image at aortic annulus level.
- Trace the perimeter of the basal annulus (Figure 9, left). Place cross-hairs at site of basal annulus, create major diameter through the site, create minor diameter defined as perpendicular to major and through site (Figure 9, right).



Figure 9. Example of perimeter measurement (left) and major and minor diameter measurements (right).

#### Sinus of Valsalva measurements

Choose the best diastolic images for measurement of sinus of Valsalva diameters and heights from images using the same reformatting technique as described in section "Reformatting of Images."

### Sinus of Valsalva diameters

- Select the double oblique axial image where the widest portion of the three sinuses is visible.
- Measure a diameter from each commissure through the site of the root to the opposite sinus. Complete for all three sinuses (Figure 3).






Figure 30. Example of sinus of Valsalva diameters

### Sinus of Valsalva heights

- The sinotubular junction is typically not co-planar with the aortic annulus. Therefore, a sinus of Valsalva height must be measured for each of the three sinuses. This height is defined as the distance between the aortic annular plane and the tallest point in the sinus.
- Choose the double oblique axial image so that it is located at the level of the aortic annulus. The reformatting line representing the double oblique axial image should now be visible in the oblique coronal and oblique sagittal images at the level of the aortic annulus.
- For the left coronary and non-coronary heights, use the oblique coronal image. For the right coronary height, use the oblique sagittal image.
- To complete the measurement, scroll through the oblique coronal or sagittal image (depending on which sinus you are measuring) and locate the heights location of the sinotubular junction. On that image, measure the distance along the path of the aortic root from the aortic annular plane, marked by the reformatting line, to the sinotubular junction (Figure 11).










Figure 41. Examples of sinus of Valsalva heights; (A) left coronary; (B) non-coronary; (C) right coronary

## 19.4.3 Anatomic suitability and valve size selection

| | Aortic annulus | | Sinus of Valsalva | |
|---|---|---|---|---|
| Device size | Perimeter<br>(mm) | Mean diameter<br>(mm) | Mean diameter<br>(mm) | Mean height<br>(mm) |
| 23 mm | 56.5 – 62.8 | 18-20 | ≥ 25 | ≥15 |
| 26 mm | 62.8 – 72.3 | 20 – 23 | ≥ 27 | ≥15 |
| 29 mm | 72.3 – 81.6 | 23 – 26 | ≥ 29 | ≥15 |

## 19.5 Resheath and Recapture Definitions

The following definitions are applicable to the data elements on the Implant e-CRF that address the use of the resheath and recapture feature.

| Resheath<br>attempt | An attempt to intentionally resheath only a portion of the Evolut™ PRO or Evolut™ PRO+ TAV (including the frame) into the capsule of the delivery catheter (e.g. with the intent to reposition of the valve during deployment). |
|---|---|
| Recapture<br>attempt | An attempt to intentionally fully resheath the entire Evolut™ PRO or Evolut™ PRO+ TAV (including the frame) into the capsule of the delivery catheter until there is no gap between capsule and the tip (e.g. with the intent to enable re-crossing of the aortic valve or retrieval of the system). |






# **19.6 Endpoint Definitions**

| Mortality | |
|---|---|
| Cardiovascular | Any of the following criteria: |
| mortality | <ol> <li>Death due to proximate cardiac cause (e.g. myocardial infarction, cardiac tamponade, worsening heart failure)</li> <li>Death caused by non-coronary vascular conditions such as neurological</li> </ol> |
| | events, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular disease |
| | <ol> <li>All procedure-related deaths, including those related to a complication of the<br/>procedure or treatment for a complication of the procedure</li> </ol> |
| | 4) All valve-related deaths including structural or nonstructural valve dysfunction or other valve-related adverse events |
| | 5) Sudden or unwitnessed death |
| | 6) Death of unknown cause |
| Non-cardiovascular mortality | Any death in which the primary cause of death is clearly related to another condition (e.g. trauma, cancer, suicide). |

| Myocardial Infarction | |
|---|---|
| Periprocedural MI<br>(≤72 h after the<br>index procedure) | New ischemic symptoms (e.g. chest pain or shortness of breath), or new ischemic signs (e.g. ventricular arrhythmias, new or worsening heart failure, new ST-segment changes, hemodynamic instability, new pathological Q-waves in at least 2 contiguous leads, imaging evidence of new loss of viable myocardium or new wall motion abnormality) AND Elevated cardiac biomarkers (preferable CK-MB) within 72 h after the index procedure, consisting of at least 1 sample post procedure with a peak value exceeding 15x as the upper reference limit for troponin or 5x for CK-MB. If cardiac biomarkers are increased at baseline (>99th percentile), a further increase in at least 50% post procedure is required AND the peak value must exceed the previously stated limit. |
| Spontaneous MI<br>(>72 h after the<br>index procedure) | Any of the following criteria: Detection of rise and/or fall of cardiac biomarkers (preferably troponin) with at least 1 value above the 99th percentile URL, together with the evidence of myocardial ischemia with at least 1 of the following: • Symptoms of ischemia |




- ECG changes indicative of new ischemia [new ST-T changes or new left bundle branch block (LBBB)]
- New pathological Q-waves in at least 2 contiguous leads
- Imaging evidence of a new loss of viable myocardium or new wall motion abnormality
- Sudden, unexpected cardiac death, involving cardiac arrest, often with symptoms suggestive of myocardial ischemia, and accompanied by presumably new ST elevation, or new LBBB, and/or evidence of fresh thrombus by angiography and/or at autopsy, but death occurring before blood samples could be obtained, or at a time before the appearance of cardiac biomarkers in the blood.
- Pathological findings of an acute myocardial infarction

| Stroke and TIA | |
|---|---|
| Diagnostic Criteria | <ol> <li>Acute episode of a focal or global neurological deficit with at least 1 of the following: <ul> <li>change in the level of consciousness</li> <li>hemiplegia, hemiparesis</li> <li>numbness or sensory loss affecting 1 side of the body</li> <li>dysphasia or aphasia</li> <li>hemianopia</li> <li>amaurosis fugax</li> <li>other neurological signs or symptoms consistent with stroke</li> </ul> </li> <li>Stroke: duration of a focal or global neurological deficit ≥24 h; OR &lt;24 h if available neuroimaging documents a new hemorrhage or infarct; OR the neurological deficit results in death</li> <li>TIA: duration of a focal or global neurological deficit &lt;24 h, any variable</li> </ol> |
| | neuroimaging does not demonstrate a new hemorrhage or infarct 2) No other readily identifiable non-stroke cause for the clinical presentation |
| | (e.g. brain tumor, trauma, infection, hypoglycemia, peripheral lesion, pharmacological influences), to be determined by or in conjunction with the designated neurologist |
| | <ul> <li>Confirmation of the diagnosis by at least 1 of the following:</li> <li>Neurologist or neurosurgical specialist</li> </ul> |

### Medtronic Confidential

diagnosed on clinical grounds alone

Neuroimaging procedure (CT scan or brain MRI), but stroke may be

**Disabling stroke:** an mRS score of 2 or more at 90 days and an increase in

at least 1 mRS category from an individual's pre-stroke baseline

**Stroke Definitions** 

Stroke and TIA


Medtronic

| | <ul> <li>Non-disabling stroke: an mRS score of &lt;2 at 90 days or one that does not<br/>result in an increase in at least 1 mRS category from an individual's pre-<br/>stroke baseline</li> </ul> |
|---|---|
| Stroke Classification | <ul> <li>Ischemic: an acute episode of focal cerebral, spinal, or retinal<br/>dysfunction caused by infarction of the central nervous system tissue</li> </ul> |
| | <ul> <li>Hemorrhagic: an acute episode of focal or global cerebral or spinal<br/>dysfunction caused by intraparenchymal, intraventricular, or<br/>subarachnoid hemorrhage</li> </ul> |
| | <ul> <li>Undetermined: insufficient information to allow categorization as<br/>ischemic or hemorrhagic</li> </ul> |

| Signs and Symptoms of Aortic Valve Disease | |
|---|---|
| Sign/Symptom | Definition |
| Aortic Valve Dysfunction | |
| Shortness of breath/dyspnea | A feeling of difficult or labored breathing that is out of |
| | proportion to the patient's level of physical activity |
| Exercise intolerance | A condition where the patient is unable to do physical exercise |
| | at the level or for the duration that would be expected of |
| | someone in his/her general physical condition, or experiences |
| | unusually severe post-exercise pain, fatigue, or other negative |
| | effects |
| Dizziness/syncope | Lightheadness or unsteadiness of gait or a partial or complete |
| | loss of consciousness with interruption of awareness of |
| | oneself and ones surroundings |
| Chest pain | Discomfort and soreness in and around the chest |
| Worsening Heart Failure | |
| Volume Overload | |
| Orthopnea | Dyspnea in which the person can breathe comfortably only |
| | when standing or sitting erect |
| Paroxysmal nocturnal dyspnea | Acute dyspnea caused by the lung congestion and edema that |
| | results from partial heart failure and occurring suddenly at |
| | night, usually an hour or two after the individual has fallen |
| | asleep. |
| Jugular venous distension | With the patient is positioned under 45°, and the filling level of |
| | the jugular vein determined. An abnormal response is more |
| | than 3 centimeters above the sternal angle. |




| Hepatomegaly | Palpation of the edge of the liver below the edge of the ribs |
|---|---|
| | without inspiration |
| Peripheral edema | Swelling of tissues, usually in the lower limbs, due to the |
| | accumulation of fluids. |
| Pulmonary rales | Small clicking, bubbling, or rattling sounds in the lung |
| | associated with inspiration |
| Abdominal-jugular reflux | An elevation of venous pressure visible in the jugular veins and |
| | measurable in the veins of the arm, produced in active or |
| | impending congestive heart failure by firm pressure with the |
| | flat hand over the abdomen. |
| Radiographic evidence of pulmonary | NA |
| edema | |
| Elevated B-type natriuretic peptide | NA |
| level | |
| Hypoperfusion | |
| Narrow pulse pressure | Pulse pressure < 30 mmHg |
| Hypotension | Systolic BP < 90 systolic |
| Renal or hepatic dysfunction | Rise in baseline creatinine by 25% |
| | <ul> <li>Increase in LFT (SGOT, SGPT) &gt; 2 times normal</li> </ul> |
| Low serum sodium concentration | Serum sodium < 130 mEq/dL |

| Bleeding Complicatio | Bleeding Complications |
|---|---|
| Life-threatening or disabling bleeding | <ul> <li>Fatal bleeding (BARC type 5) OR</li> <li>Bleeding in a critical organ, such as intracranial, intraspinal,</li> <li>intraocular, or pericardial necessitating pericardiocentesis, or intramuscular with compartment syndrome (BARC type 3b and 3c) OR</li> <li>Bleeding causing hypovolemic shock or severe hypotension requiring vasopressors or surgery (BARC type 3b) OR</li> <li>Overt source of bleeding with drop in hemoglobin ≥5 g/dL or whole blood</li> </ul> |
| | or packed red blood cells (RBCs) transfusion ≥4 units* (BARC type 3b) |
| Major bleeding (BARC type 3a) | <ol> <li>Overt bleeding either associated with a drop in the hemoglobin level of at least 3.0 g/dL or requiring transfusion of 2 or 3 units of whole blood/RBC, or causing hospitalization or permanent injury, or requiring surgery AND</li> <li>Does not meet criteria of life-threatening or disabling bleeding</li> </ol> |
| Minor bleeding | Any bleeding worthy of clinical mention (e.g. access site hematoma) that |
| (BARC type 2 or | does not qualify as life-threatening, disabling, or major |




| 3a, depending |
|------------------|
| on the severity) |

\*Given one unit of packed RBC typically will raise hemoglobin concentration by 1 g/dL, an estimated decrease in hemoglobin will be calculated; BARC: Bleeding Academic Research Consortium; RBC: red blood cell

#### Notes:

- 1. With respect to blood transfusions, it is critical to acknowledge that a bleeding complication has to be the result of overt bleeding and cannot be adjudicated based on blood transfusions alone.
- 2. Pre-operative hemoglobin will be used to determine severity of bleeding events

| Acute Kidney Injury (up to 7 days post procedure) | |
|---|---|
| Stage 1 | <ol> <li>Increase in serum creatinine to 150%-199% (1.5-1.99 x increase compared with baseline) OR increase of ≥0.3 mg/dL (≥26.4 mmol/L) OR</li> <li>Urine output &lt;0.5 mL/kg/h for &gt;6 but &lt;12 h</li> </ol> |
| Stage 2 | <ol> <li>Increase in serum creatinine to 200%-299% (2.0%-2.99% increase compared with baseline) OR</li> <li>Urine output &lt;0.5 mL/kg/h for &gt;12 but &lt;24 h</li> </ol> |
| Stage 3 | <ol> <li>Increase in serum creatinine to ≥300% (&gt;3 x increase compared with baseline) OR serum creatinine of ≥4.0 mg/dL (≥354 mmol/L) with an acute increase of at least 0.5 mg/dL (44 mmol/L) OR</li> <li>Urine output &lt;0.3 ml/kg/h for ≥24 h OR</li> <li>Anuria for ≥12 h</li> </ol> |

| Vascular Access Site a | nd A | ccess Related Complications |
|---|---|---|
| Major vascular complication | 1) | Any aortic dissection, aortic rupture, annulus rupture, left ventricle perforation, or new apical aneurysm/pseudoaneurysm OR Access site or access-related vascular injury (dissection, stenosis, perforation, rupture, arterio-venous fistula, pseudoaneurysm, hematoma, irreversible nerve injury, compartment syndrome, percutaneous closure device failure) |
| | | <i>leading to</i> death, life-threatening or major bleeding, visceral ischemia, or neurological impairment OR |
| | 3) | Distal embolization (noncerebral) from a vascular source requiring surgery or resulting in amputation or irreversible end-organ damage OR |
| | 4) | The use of unplanned endovascular or surgical intervention associated with death, major bleeding, visceral ischemia or neurological impairment OR |
| | 5) | Any new ipsilateral lower extremity ischemia documented by patient symptoms, physical exam, and/or decreased or absent blood flow on lower extremity angiogram OR |
| | 6) | Surgery for access site-related nerve injury OR |




| | 7) Permanent access site-related nerve injury |
|---|---|
| Minor vascular complication | <ol> <li>Access site or access-related vascular injury (dissection, stenosis, perforation, rupture, arterio-venous fistula, pseudoaneurysms, hematomas, percutaneous closure device failure) not leading to death, life-threatening or major bleeding*, visceral ischemia, or neurological impairment OR</li> <li>Distal embolization treated with embolectomy and/or thrombectomy and not resulting in amputation or irreversible end-organ damage OR</li> <li>Any unplanned endovascular stenting or unplanned surgical intervention not meeting the criteria for a major vascular complication OR</li> <li>Vascular repair or the need for vascular repair (via surgery, ultrasound-guided compression, transcatheter embolization, or stent-graft)</li> </ol> |
| Percutaneous Closure device failure | Failure of a closure device to achieve hemostasis at the arteriotomy site leading to alternative treatment (other than manual compression or adjunctive endovascular ballooning) |

Note: Refer to VARC-2 bleeding definitions

### **Valve Dysfunction Requiring Repeat Procedure**

Any valve dysfunction that requires repeat procedure (e.g. balloon valvuloplasty, TAVR, or surgical AVR)

Note: Repeat procedures are reported on the appropriate e-CRF

| Other TAVR Related Complications | |
|---|---|
| Conversion to open surgery | Conversion to open sternotomy during the TAVR procedure secondary to any procedure-related complications Conversions to open surgery will be considered serious adverse events |
| Unplanned use of cardiopulmonary bypass | regardless of reason for the surgical conversion. Unplanned use of CPB for hemodynamic support at any time during the TAVR procedure |
| Coronary artery obstruction | Angiographic or echocardiographic evidence of a new, partial or complete, obstruction of a coronary ostium, either by the Evolut™ PRO prosthesis itself, the native leaflets, calcifications, or dissection, occurring during or after the TAVR procedure. |
| Ventricular septal perforation | Angiographic or echocardiographic evidence of a new septal perforation during or after the TAVR procedure |
| Mitral valve<br>apparatus damage<br>or dysfunction | Angiographic or echocardiographic evidence of new damage (chordae, papillary muscle, or leaflet) to the mitral valve apparatus or dysfunction (e.g. restrictions due to the Evolut™ PRO) of the mitral valve during or after the TAVR procedure |




| Cardiac tamponade | Evidence of new pericardial effusion associated with hemodynamic instability and clearly related to the TAVR procedure |
|---|---|
| Valve Thrombosis<br>(Clinical) | Any thrombus not caused by infection attached to or near the trial valve that occludes part of the blood flow path, interferes with valve function, or is sufficiently large to warrant treatment which is associated with any of the following clinical sequelae.: • Thromboembolic complications including |
| | <ul> <li>Any ischemic stroke</li> </ul> |
| | <ul> <li>Any peripheral embolic event</li> </ul> |
| | <ul> <li>ST segment elevation or Non-ST elevation myocardial infarction</li> </ul> |
| | Hemodynamic impairment associated with a worsening of heart failure |
| | Note: valve thrombus found at autopsy in a subject whose cause of death was not valve-related or found at operation for an unrelated indication should not be reported as valve thrombosis |
| Valve Thrombosis<br>(Sub-Clinical) | Any thrombus not caused by infection attached to or near the trial valve that occludes part of the blood flow path or interferes with valve function, without evident clinical sequelae, causing a hemodynamic impediment meeting the following criteria: • Increase in aortic regurgitation to moderate to severe. |
| | An increase by more than 50% of discharge mean aortic valve gradient (with the post discharge mean gradient being ≥ 20 mmHg) or a decrease in the Doppler Velocity Index (DVI) by more than 50% |
| Leaflet Motion | Possible leaflet motion abnormality identified by any imaging modality with |
| Abnormality (With | medical therapy (e.g. anticoagulation therapy, fibrinolytic therapy or valve- |
| Treatment) | related medical intervention) initiated and without significant negative |
| | change in valve function (i.e. increasing obstruction or central regurgitation). |
| Leaflet Motion | Possible leaflet motion abnormality identified by any imaging modality |
| | without medical therapy (e.g. anticoagulation therapy, fibrinolytic therapy |
| Abnormality | or valve-related medical intervention) initiated but without significant |
| (Without | negative change in valve function (i.e. increasing obstruction or central |
| Treatment) | regurgitation). |
| Valve migration | After initial correct positioning, any observed movement (upward or downward) of the Evolut™ PRO within the aortic annulus from its initial position, with or without consequences. |
| Valve embolization | The Evolut™ PRO moves during or after deployment such that it loses contact within the aortic annulus* |




| Ectopic valve | Permanent deployment of the Evolut™ PRO in a location other than the aortic |
|---|---|
| deployment | root |
| Valve in Valve<br>deployment | Additional valve prosthesis is implanted within a previously implanted Evolut™ PRO because of sub-optimal device position and/or function, during or after the index procedure. |
| Hemolysis | Red cell destruction as evidenced by plasma free hemoglobin >50 mg/dl |
| | Minor hemolysis: No intervention required Major hemolysis: Requires intervention (e.g. iron supplements, transfusion, invasive intervention). |
| Frame fracture | Visual evidence on radiography or at explant of loss of contact between elements (cells) of the stent. |
| | <b>Minor frame fracture:</b> Does not require intervention or is not associated with prosthetic valve dysfunction. |
| | Major frame fracture: Intervention required (e.g. reoperation, catheter reintervention) or is associated with prosthetic valve dysfunction |
| TAVR Conversion to Other Percutaneous Procedure | Any conversion of the intended TAVR procedure, prior to closure to other percutaneous intervention due to technical challenges, technical contraindications to the intended procedure identified intra-procedurally or complications. |
| Aborted Procedure | Termination of the procedure prior to implantation of the valve due to identification of a technical contraindication, intraprocedural complications of a concomitant procedure prior to valve implantation or radiation dosage. Aborted procedures will be considered serious adverse events regardless of reason for termination of the procedure. |
| Reintervention –<br>Surgical or<br>Percutaneous | Any surgical or percutaneous interventional catheter procedure that repairs, otherwise alters or adjusts, or replaces a previously implanted valve. In addition to surgical reoperations, balloon dilatation, interventional manipulation, repositioning, or retrieval, and other catheter-based interventions for valve-related complications are also considered reinterventions. Reintervention is further subdivided into surgical and percutaneous. Relationship to the study valve will be assessed for the most current valve implanted or attempted to be implanted. |

<sup>\*</sup>Valve embolizations are not applicable to valve that move during the procedure but are able to be recaptured and repositioned.

### **Prosthetic Valve Endocarditis**


Page 88 of 89



### Any of the following:

- 1) Fulfillment of the following Duke criteria (22) for definite endocarditis:
  - Histologic and/or microbiologic evidence of infection at surgery or autopsy, or
  - 2 major criteria, or
  - 1 major criteria or 3 minor criteria, or
  - 5 minor criteria

Major and minor criteria are as follows:

#### **Major Criteria**:

- Blood cultures positive for Infective Endocarditis (IE)
  - Typical microorganisms consistent with IE isolated from two separate blood cultures, as noted below
    - Viridans streptococci, Streptococcus bovis, Staphylcoccus aureus, or HACEK group
    - Community-acquired enterococci in the presence of a primary focus
  - Microorganisms consistent with IE isolated from persistently positive blood cultures defined as:
    - At least two positive cultures or blood samples obtained >12 hours apart, or
    - All of three, or a majority of four or more separate cultures of blood, the first and last sample obtained > one hour apart
  - Single blood culture positive for Coxiella burnetti or an antiphase I IG antibody titer >1:800
- · Evidence of endocardial involvement
  - Positive results of echocardiography for IE defined as:
    - Oscillating intracardiac mass on a valve or supporting structures in the path of regurgitant jets or on implanted material in the absence of an anatomic explantation, or
    - Abscess, or
    - New partial dehiscence of a valvular prosthesis
  - New valvular regurgitation (worsening or changing or pre-existing murmur not sufficient)

#### **Minor Criteria:**

- Predisposition: predisposing heart condition or intravenous drug use
- Fever: temperature >38°C
- Vascular phenomena: major arterial emboli, septic pulmonary infarcts, mycotic aneurysm, intracranial hemorrhage, conjunctival hemorrhages, and Janeway's lesions
- Immunological phenomena: glomerulonephritis, Osler's nodes, Roth's spots, and rheumatoid factor
- Microbiological evidence: positive blood culture but does not meet a major criterion (as noted above) or serological evidence of active infection with organism consistent with infectious endocarditis.
- Echocardiographic findings: consistent with IE but do not meet a major criterion as noted

If only 1 major and 1-2 minor criteria are fulfilled, or if only 3-4 minor criteria are fulfilled, the



Page 89 of 89



event will be coded as "possible endocarditis"

- 2) Evidence of abscess, paravalvular leak, pus, or vegetation confirmed as secondary to infection by histological or bacteriological studies during a re-operation
- 3) Findings of abscess, pus, or vegetation involving the Evolut™ PRO at autopsy

| Prosthetic Valve Dysfunction | |
|---|---|
| Stenosis: mild | For subjects with BSA $\geq$ 1.6 m <sup>2</sup> : Mean aortic gradient $\geq$ 20 and $\leq$ 40 mmHg, EOA $\geq$ 0.8 and $\leq$ 1.1 cm <sup>2</sup> AND/OR DVI $\geq$ 0.25 and $\leq$ 0.35 For subjects with BSA $<$ 1.6 m <sup>2</sup> : Mean aortic gradient $\geq$ 20 and $\leq$ 40 mmHg, EOA $\geq$ 0.6 cm <sup>2</sup> and $\leq$ 0.9 cm <sup>2</sup> AND/OR DVI $\geq$ 0.25 and $\leq$ 0.35 |
| Stenosis: moderate/severe | For subjects with BSA ≥ 1.6 m <sup>2</sup> : Mean aortic gradient > 40 mmHg, EOA < 0.8 cm <sup>2</sup> AND/OR DVI < 0.25 For subjects with BSA < 1.6 m <sup>2</sup> : Mean aortic gradient > 40 mmHg, EOA < 0.6 cm <sup>2</sup> AND/OR DVI < 0.25 |
| Paravalvular regurgitation: moderate | Moderate paravalvular regurgitation (per echo criteria in CIP) |
| Paravalvular regurgitation: severe | Severe paravalvular regurgitation (per echo criteria in CIP) |
| Transvalvular regurgitation: moderate | Moderate transvalvular regurgitation (per echo criteria in CIP) |
| Transvalvular regurgitation: severe | Severe transvalvular regurgitation (per echo criteria in CIP) |

#### Notes:

- DVI = Doppler Velocity Index (LVOT VTI/valve VTI)
- For subjects LVOT diameter > 2.5 cm, the DVI criteria for significant (moderate or severe) stenosis is 0.2
- Reporting of prosthetic valve dysfunction will be based on core lab values (if available).
- Prosthetic valve dysfunction events are not reported as adverse events, unless the dysfunction is
  accompanied with clinical sequelae at the time of event detection, and the clinical sequelae are
  chronologically and physiologically associated with the dysfunction. However, prosthetic
  dysfunctions that are associated with adverse events, and that meet the definition of a serious
  adverse event, should be reported as such.